CLINICAL TRIAL: NCT03110107
Title: Phase 1/2a First-In-Human Study of BMS-986218 Monoclonal Antibody Alone and in Combination With Nivolumab in Advanced Solid Tumors
Brief Title: First-In-Human Study of Monoclonal Antibody BMS-986218 by Itself and in Combination With Nivolumab in Participants With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business Objectives have changed.
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA022-001; 2017-000597-11 (EudraCT Number)
Record Dates: First submitted 2017-04-07; First posted 2017-04-12 (Actual); Results first posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Advanced Cancer
Keywords: BMS-986218; Nivolumab; Ipilimumab
MeSH Terms: interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1A: Monotherapy (BMS-986218) (Experimental)
  Interventions: Biological: BMS-986218
- Part 1B: Combination Therapy (BMS-986218 + Nivolumab) (Experimental)
  Interventions: Biological: BMS-986218; Biological: Nivolumab
- Part 2A: Monotherapy (BMS-986218 OR Ipilimumab) (Experimental)
  Interventions: Biological: Ipilimumab; Biological: BMS-986218
- Part 2B: Monotherapy (BMS-986218) (Experimental)
  Interventions: Biological: BMS-986218
- Part 2C: Expansion Combination Therapy (BMS-986218 + Nivolumab) (Experimental)
  Interventions: Biological: BMS-986218; Biological: Nivolumab
- Part 2D: Expansion Combination Therapy (BMS-986218 + Nivolumab) (Experimental)
  Interventions: Biological: BMS-986218; Biological: Nivolumab

INTERVENTIONS:
Biological: Ipilimumab — Specified dose on specified days
  Other Names: Yervoy
  Arms: Part 2A: Monotherapy (BMS-986218 OR Ipilimumab)
Biological: BMS-986218 — Specified dose on specified days
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo
  Arms: Part 1B: Combination Therapy (BMS-986218 + Nivolumab); Part 2C: Expansion Combination Therapy (BMS-986218 + Nivolumab); Part 2D: Expansion Combination Therapy (BMS-986218 + Nivolumab)

SUMMARY:
The purpose of this study is to determine whether BMS-986218 both by itself and in combination with Nivolumab is safe and tolerable in the treatment of advanced solid tumors.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Histologic or cytologic confirmation of a solid tumor that is advanced (metastatic, recurrent and/or unresectable)
* Eastern Cooperative Oncology Group Performance Status of 0 or 1
* Participants must have received, and then progressed, relapsed, or been intolerant to at least 2 standard treatment regimens with proven survival benefit in the advanced or metastatic setting according to tumor type, if such a therapy exists
* Advanced stage cutaneous melanoma who have received standard therapies with proven survival benefit including prior immunotherapy with an anti-programmed cell death 1 (anti-PD-1) or anti-programmed death ligand 1 (anti-PD-L1) (For Part 2A)
* Non-small cell lung cancer (NSCLC) (adenocarcinoma or squamous cell carcinoma) who have received standard therapies with proven survival benefit including prior immunotherapy with an anti-PD-1 or anti-PD-L1 (For Parts 2B & 2C)
* Microsatellite Stable Colorectal Cancer (MSS CRC) who have received standard therapies with proven survival benefit (Part 2D)

Exclusion Criteria:

* Participants with primary CNS malignancies, or tumors with CNS metastases as the only site of disease, will be excluded
* Cytotoxic agents, unless at least 4 weeks have elapsed from last dose of prior anti-cancer therapy and initiation of study therapy
* Prior anti-cancer treatments such as chemotherapy, radiotherapy, hormonal, or immunotherapy (including anti-PD-1/PD-L1) are permitted

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (52):
- United States (9):
  - Local Institution - 0058, Atlanta, Georgia
  - Local Institution - 0025, Boston, Massachusetts
  - Local Institution - 0002, Hackensack, New Jersey
  - Local Institution - 0028, New Brunswick, New Jersey
  - Local Institution - 0001, New York, New York
  - Local Institution - 0007, New York, New York
  - Local Institution - 0015, Monroeville, Pennsylvania
  - Local Institution - 0004, Philadelphia, Pennsylvania
  - Local Institution - 0033, Sioux Falls, South Dakota
- Argentina (7):
  - Local Institution - 0042, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 0053, ABB, Buenos Aires F.D.
  - Local Institution - 0057, CABA, Buenos Aires F.D.
  - Local Institution - 0062, Córdoba, Córdoba Province
  - Local Institution - 0060, Río Cuarto, Córdoba Province
  - Local Institution - 0047, Villa Siburu, Córdoba Province
  - Local Institution - 0059, Buenos Aires, Distrito Federal
- Australia (3):
  - Local Institution - 0026, Northmead, New South Wales
  - Local Institution - 0006, Wollstonecraft, New South Wales
  - Local Institution - 0049, Murdoch, Western Australia
- Local Institution - 0039, Ghent, Belgium
- Canada (4):
  - Local Institution - 0037, Edmonton, Alberta
  - Local Institution - 0023, Vancouver, British Columbia
  - Local Institution - 0027, Ottawa, Ontario
  - Local Institution - 0022, Toronto, Ontario
- Chile (3):
  - Local Institution - 0052, Viña del Mar, Región de Valparaíso
  - Local Institution - 0048, Santiago, Santiago Metropolitan
  - Local Institution - 0041, Santiago, Santiago Metropolitan
- Local Institution - 0045, Helsinki, Finland
- France (3):
  - Local Institution - 0019, Lyon
  - Local Institution - 0020, Toulouse
  - Local Institution - 0018, Villejuif
- Germany (2):
  - Local Institution - 0009, Dresden
  - Local Institution - 0030, Essen
- Israel (2):
  - Local Institution - 0029, Haifa
  - Local Institution - 0008, Ramat Gan
- Italy (3):
  - Local Institution - 0011, Napoli
  - Local Institution - 0061, Rozzano
  - Local Institution - 0010, Siena
- Netherlands (2):
  - Local Institution - 0038, Amsterdam
  - Local Institution - 0043, Nijmegen
- Local Institution - 0040, Oslo, Norway
- Local Institution - 0036, Warsaw, Poland
- Romania (2):
  - Local Institution - 0034, Cluj-Napoca
  - Local Institution - 0035, Craiova
- Spain (6):
  - Local Institution - 0014, Barcelona
  - Local Institution - 0056, Madrid
  - Local Institution - 0055, Madrid
  - Local Institution - 0013, Madrid
  - Local Institution - 0054, Málaga
  - Local Institution - 0012, Pamplona
- Switzerland (2):
  - Local Institution - 0017, Lausanne
  - Local Institution - 0031, Zurich

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/home

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part 1, Part 2C and Part 2D were non-randomized. Part 2A and Part 2B were randomized.
Groups:
- Part 1A: BMS-986218 2 mg All Solid Tumors: Participants received BMS-986218 at 2 mg every 4 weeks for up to 2 years
- Part 1A: BMS-986218 4 mg All Solid Tumors: Participants received BMS-986218 at 4 mg every 4 weeks for up to 2 years
- Part 1A: BMS-986218 7 mg All Solid Tumors: Participants received BMS-986218 at 7 mg every 4 weeks for up to 2 years
- Part 1A: BMS-986218 20 mg All Solid Tumors: Participants received BMS-986218 at 20 mg every 4 weeks for up to 2 years
- Part 1A: BMS-986218 40 mg All Solid Tumors: Participants received BMS-986218 at 40 mg every 4 weeks for up to 2 years
- Part 1A: BMS-986218 70 mg All Solid Tumors: Participants received BMS-986218 at 70 mg every 4 weeks for up to 2 years
- Part 1A: BMS-986218 100 mg All Solid Tumors: Participants received BMS-986218 at 100 mg every 4 weeks for up to 2 years
- Part 1A: BMS-986218 150 mg All Solid Tumors: Participants received BMS-986218 at 150 mg every 4 weeks for up to 2 years
- Part 1A: BMS-986218 200 mg All Solid Tumors: Participants received BMS-986218 at 200 mg every 4 weeks for up to 2 years
- Part 1A: BMS-986218 20 mg Select Solid Tumors: Participants received BMS-986218 at 20 mg every 2 weeks for up to 2 years
- Part 1A: BMS-986218 35 mg Select Solid Tumors: Participants received BMS-986218 at 35 mg every 2 weeks for up to 2 years
- Part 1A: BMS-986218 50 mg Select Solid Tumors: Participants received BMS-986218 at 50 mg every 2 weeks for up to 2 years
- Part 1A: BMS-986218 20 mg Select Solid Tumors Pharmacodynamics Cohort: Participants received BMS-986218 at 20 mg every 2 weeks
- Part 1B: BMS-986218 7 mg + Nivolumab 480 mg Select Solid Tumors: Participants received BMS-986218 at 7 mg with nivolumab at 480 mg every 4 weeks
- Part 1B: BMS-986218 20 mg + Nivolumab 480 mg Select Solid Tumors: Participants received BMS-986218 at 20 mg with nivolumab at 480 mg every 4 weeks
- Part 1B: BMS-986218 40 mg + Nivolumab 480 mg Select Solid Tumors; Part 2C: BMS-986218 + Nivolumab Non-Small Cell Lung Cancer (NSCLC); Part 2D: BMS-986218 + Nivolumab Microsatellite Stable Colorectal Cancer (MSS CRC): Participants received BMS-986218 at 40 mg with nivolumab at 480 mg every 4 weeks
- Part 1B: BMS-986218 70 mg + Nivolumab 480 mg Select Solid Tumors: Participants received BMS-986218 at 70 mg with nivolumab at 480 mg every 4 weeks
- Part 2A: Ipilimumab Cutaneous Melanoma: Participants received ipilimumab at 3 mg/kg every 3 weeks
- Part 2A: BMS-986218 7 mg Cutaneous Melanoma; Part 2B: BMS-986218 7 mg Non-Small Cell Lung Cancer (NSCLC): Participants received BMS-986218 at 7 mg every 4 weeks
- Part 2A: BMS-986218 20 mg Cutaneous Melanoma; Part 2B: BMS-986218 20 mg Non-Small Cell Lung Cancer (NSCLC): Participants received BMS-986218 at 20 mg every 4 weeks
- Part 2A: BMS-986218 70 mg Cutaneous Melanoma; Part 2B: BMS-986218 70 mg Non-Small Cell Lung Cancer (NSCLC): Participants received BMS-986218 at 70 mg every 4 weeks
Period: Pre-treatment Period
Arm/Group | Part 1A: BMS-986218 2 mg All Solid Tumors | Part 1A: BMS-986218 4 mg All Solid Tumors | Part 1A: BMS-986218 7 mg All Solid Tumors | Part 1A: BMS-986218 20 mg All Solid Tumors | Part 1A: BMS-986218 40 mg All Solid Tumors | Part 1A: BMS-986218 70 mg All Solid Tumors | Part 1A: BMS-986218 100 mg All Solid Tumors | Part 1A: BMS-986218 150 mg All Solid Tumors | Part 1A: BMS-986218 200 mg All Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors | Part 1A: BMS-986218 35 mg Select Solid Tumors | Part 1A: BMS-986218 50 mg Select Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors Pharmacodynamics Cohort | Part 1B: BMS-986218 7 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 20 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 40 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 70 mg + Nivolumab 480 mg Select Solid Tumors | Part 2A: Ipilimumab Cutaneous Melanoma | Part 2A: BMS-986218 7 mg Cutaneous Melanoma | Part 2A: BMS-986218 20 mg Cutaneous Melanoma | Part 2A: BMS-986218 70 mg Cutaneous Melanoma | Part 2B: BMS-986218 7 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 20 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 70 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2C: BMS-986218 + Nivolumab Non-Small Cell Lung Cancer (NSCLC) | Part 2D: BMS-986218 + Nivolumab Microsatellite Stable Colorectal Cancer (MSS CRC)
Started (Randomized) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 19 | 18 | 18 | 22 | 22 | 22 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 19 | 18 | 18 | 22 | 22 | 22 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period
Arm/Group | Part 1A: BMS-986218 2 mg All Solid Tumors | Part 1A: BMS-986218 4 mg All Solid Tumors | Part 1A: BMS-986218 7 mg All Solid Tumors | Part 1A: BMS-986218 20 mg All Solid Tumors | Part 1A: BMS-986218 40 mg All Solid Tumors | Part 1A: BMS-986218 70 mg All Solid Tumors | Part 1A: BMS-986218 100 mg All Solid Tumors | Part 1A: BMS-986218 150 mg All Solid Tumors | Part 1A: BMS-986218 200 mg All Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors | Part 1A: BMS-986218 35 mg Select Solid Tumors | Part 1A: BMS-986218 50 mg Select Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors Pharmacodynamics Cohort | Part 1B: BMS-986218 7 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 20 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 40 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 70 mg + Nivolumab 480 mg Select Solid Tumors | Part 2A: Ipilimumab Cutaneous Melanoma | Part 2A: BMS-986218 7 mg Cutaneous Melanoma | Part 2A: BMS-986218 20 mg Cutaneous Melanoma | Part 2A: BMS-986218 70 mg Cutaneous Melanoma | Part 2B: BMS-986218 7 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 20 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 70 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2C: BMS-986218 + Nivolumab Non-Small Cell Lung Cancer (NSCLC) | Part 2D: BMS-986218 + Nivolumab Microsatellite Stable Colorectal Cancer (MSS CRC)
Started (Treated) | 4 | 9 | 12 | 15 | 12 | 14 | 7 | 11 | 5 | 14 | 6 | 4 | 1 | 5 | 17 | 19 | 7 | 20 | 19 | 18 | 18 | 22 | 22 | 22 | 29 | 44
Completed | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 13 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Not Completed | 4 | 9 | 12 | 14 | 12 | 13 | 7 | 11 | 5 | 14 | 6 | 4 | 1 | 5 | 16 | 19 | 7 | 7 | 19 | 18 | 18 | 20 | 22 | 22 | 29 | 43
Not completed — Disease Progression | 3 | 9 | 8 | 11 | 8 | 4 | 6 | 7 | 2 | 10 | 5 | 2 | 0 | 5 | 14 | 14 | 4 | 3 | 16 | 14 | 12 | 16 | 18 | 13 | 16 | 31
Not completed — Study drug toxicity | 1 | 0 | 1 | 2 | 0 | 3 | 1 | 1 | 3 | 2 | 0 | 2 | 0 | 0 | 2 | 3 | 3 | 3 | 1 | 2 | 2 | 0 | 2 | 6 | 7 | 6
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 1 | 4 | 2 | 2 | 2 | 2 | 4
Not completed — Participant request to discontinue study treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Participant withdrew consent | 0 | 0 | 1 | 0 | 4 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 2
Not completed — Participants no longer meets study criteria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other Reasons | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1A: BMS-986218 2 mg All Solid Tumors | Part 1A: BMS-986218 4 mg All Solid Tumors | Part 1A: BMS-986218 7 mg All Solid Tumors | Part 1A: BMS-986218 20 mg All Solid Tumors | Part 1A: BMS-986218 40 mg All Solid Tumors | Part 1A: BMS-986218 70 mg All Solid Tumors | Part 1A: BMS-986218 100 mg All Solid Tumors | Part 1A: BMS-986218 150 mg All Solid Tumors | Part 1A: BMS-986218 200 mg All Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors | Part 1A: BMS-986218 35 mg Select Solid Tumors | Part 1A: BMS-986218 50 mg Select Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors Pharmacodynamics Cohort | Part 1B: BMS-986218 7 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 20 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 40 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 70 mg + Nivolumab 480 mg Select Solid Tumors | Part 2A: Ipilimumab Cutaneous Melanoma | Part 2A: BMS-986218 7 mg Cutaneous Melanoma | Part 2A: BMS-986218 20 mg Cutaneous Melanoma | Part 2A: BMS-986218 70 mg Cutaneous Melanoma | Part 2B: BMS-986218 7 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 20 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 70 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2C: BMS-986218 + Nivolumab Non-Small Cell Lung Cancer (NSCLC) | Part 2D: BMS-986218 + Nivolumab Microsatellite Stable Colorectal Cancer (MSS CRC) | Total
Number analyzed (Participants) | 4 | 9 | 12 | 15 | 12 | 14 | 7 | 11 | 5 | 14 | 6 | 4 | 1 | 5 | 17 | 19 | 7 | 20 | 19 | 18 | 18 | 22 | 22 | 22 | 29 | 44 | 376
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.5 (23.1) | 63.6 (11.4) | 65.6 (11.1) | 63.3 (8.3) | 60.6 (12.1) | 55.1 (9.5) | 58.7 (6.1) | 65.5 (10.1) | 57.8 (10.2) | 60.1 (12.2) | 64.7 (6.7) | 54.5 (4.1) | 76.0 (0) | 70.4 (6.1) | 58.7 (11.3) | 61.1 (9.5) | 57.7 (9.7) | 65.6 (11.6) | 61.8 (14.4) | 65.8 (14.6) | 64.6 (13.2) | 66.0 (8.6) | 65.9 (11.2) | 62.8 (7.4) | 62.7 (9.8) | 55.3 (11.5) | 61.7 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 4 | 6 | 7 | 8 | 5 | 7 | 2 | 9 | 0 | 3 | 0 | 2 | 5 | 8 | 7 | 10 | 9 | 11 | 4 | 10 | 7 | 6 | 16 | 24 | 175
  Male | 2 | 6 | 8 | 9 | 5 | 6 | 2 | 4 | 3 | 5 | 6 | 1 | 1 | 3 | 12 | 11 | 0 | 10 | 10 | 7 | 14 | 12 | 15 | 16 | 13 | 20 | 201
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 4 | 7 | 5 | 0 | 5 | 3 | 1 | 1 | 1 | 39
  Not Hispanic or Latino | 3 | 6 | 10 | 11 | 11 | 12 | 5 | 8 | 4 | 10 | 4 | 2 | 0 | 3 | 12 | 6 | 3 | 7 | 5 | 5 | 3 | 8 | 13 | 5 | 10 | 11 | 177
  Unknown or Not Reported | 0 | 0 | 0 | 3 | 1 | 0 | 2 | 3 | 1 | 3 | 2 | 2 | 0 | 2 | 4 | 13 | 4 | 9 | 7 | 8 | 15 | 9 | 6 | 16 | 18 | 32 | 160
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Asian | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 4
  White | 3 | 9 | 9 | 15 | 10 | 9 | 7 | 10 | 4 | 13 | 6 | 4 | 0 | 5 | 13 | 18 | 6 | 20 | 19 | 18 | 18 | 22 | 21 | 21 | 29 | 42 | 351
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 2 | 0 | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Time Frame: From first dose of study medication through 100 days following last dose of study treatment (assessed for an average of 8 months up to a max of approximately 28 months)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: BMS-986218 2 mg All Solid Tumors | Part 1A: BMS-986218 4 mg All Solid Tumors | Part 1A: BMS-986218 7 mg All Solid Tumors | Part 1A: BMS-986218 20 mg All Solid Tumors | Part 1A: BMS-986218 40 mg All Solid Tumors | Part 1A: BMS-986218 70 mg All Solid Tumors | Part 1A: BMS-986218 100 mg All Solid Tumors | Part 1A: BMS-986218 150 mg All Solid Tumors | Part 1A: BMS-986218 200 mg All Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors | Part 1A: BMS-986218 35 mg Select Solid Tumors | Part 1A: BMS-986218 50 mg Select Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors Pharmacodynamics Cohort | Part 1B: BMS-986218 7 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 20 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 40 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 70 mg + Nivolumab 480 mg Select Solid Tumors | Part 2A: Ipilimumab Cutaneous Melanoma | Part 2A: BMS-986218 7 mg Cutaneous Melanoma | Part 2A: BMS-986218 20 mg Cutaneous Melanoma | Part 2A: BMS-986218 70 mg Cutaneous Melanoma | Part 2B: BMS-986218 7 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 20 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 70 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2C: BMS-986218 + Nivolumab Non-Small Cell Lung Cancer (NSCLC) | Part 2D: BMS-986218 + Nivolumab Microsatellite Stable Colorectal Cancer (MSS CRC)
Number analyzed (Participants) | 4 | 9 | 12 | 15 | 12 | 14 | 7 | 11 | 5 | 14 | 6 | 4 | 1 | 5 | 17 | 19 | 7 | 20 | 19 | 18 | 18 | 22 | 22 | 22 | 29 | 44
Participants | 4 | 9 | 11 | 15 | 12 | 14 | 7 | 11 | 5 | 13 | 6 | 4 | 1 | 5 | 17 | 19 | 7 | 18 | 19 | 15 | 17 | 21 | 22 | 22 | 29 | 44

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, and requires inpatient hospitalization or causes prolongation of existing hospitalization.
Time Frame: as for outcome 1
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: BMS-986218 2 mg All Solid Tumors | Part 1A: BMS-986218 4 mg All Solid Tumors | Part 1A: BMS-986218 7 mg All Solid Tumors | Part 1A: BMS-986218 20 mg All Solid Tumors | Part 1A: BMS-986218 40 mg All Solid Tumors | Part 1A: BMS-986218 70 mg All Solid Tumors | Part 1A: BMS-986218 100 mg All Solid Tumors | Part 1A: BMS-986218 150 mg All Solid Tumors | Part 1A: BMS-986218 200 mg All Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors | Part 1A: BMS-986218 35 mg Select Solid Tumors | Part 1A: BMS-986218 50 mg Select Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors Pharmacodynamics Cohort | Part 1B: BMS-986218 7 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 20 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 40 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 70 mg + Nivolumab 480 mg Select Solid Tumors | Part 2A: Ipilimumab Cutaneous Melanoma | Part 2A: BMS-986218 7 mg Cutaneous Melanoma | Part 2A: BMS-986218 20 mg Cutaneous Melanoma | Part 2A: BMS-986218 70 mg Cutaneous Melanoma | Part 2B: BMS-986218 7 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 20 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 70 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2C: BMS-986218 + Nivolumab Non-Small Cell Lung Cancer (NSCLC) | Part 2D: BMS-986218 + Nivolumab Microsatellite Stable Colorectal Cancer (MSS CRC)
Number analyzed (Participants) | 4 | 9 | 12 | 15 | 12 | 14 | 7 | 11 | 5 | 14 | 6 | 4 | 1 | 5 | 17 | 19 | 7 | 20 | 19 | 18 | 18 | 22 | 22 | 22 | 29 | 44
Participants | 2 | 5 | 5 | 9 | 10 | 7 | 5 | 7 | 5 | 10 | 4 | 3 | 1 | 3 | 13 | 18 | 7 | 9 | 11 | 12 | 12 | 16 | 15 | 17 | 23 | 34

3. Primary Outcome: Number of Participants With Adverse Events (AEs) Meeting Protocol-defined Dose-limiting Toxicity (DLT) Criteria
Description: Dose-Limiting Toxicities (DLTs) are effects of a treatment that are serious enough to prevent an increase in dose of that treatment.
  Grade 1=Mild, 2=Moderate, 3=Severe, 4=Life-threatening, 5=Death
  Gastrointestinal DLT:
  * Grade 2 colitis >5 days
  * Grade ≥3 diarrhea/colitis
  Hepatic DLT:
  * Grade 4 serum transaminases (AST & ALT), alkaline phosphatase (ALP), or total bilirubin elevations
  * Grade 3 serum AST, ALT, or ALP elevations lasting >5 days or with clinical symptoms or bilirubin > 2×ULN without cholestasis
  Hematologic DLT:
  * Grade 4 neutropenia ≥7 days
  * Grade 4 thrombocytopenia
  Dermatologic DLT:
  * Grade 4 rash
  * Grade 3 rash if no improvement after 1-2-week infusion delay
  Other DLTs:
  * Grade 2 drug-related uveitis, episcleritis, iritis, eye pain, or blurred vision that doesn't respond to treatment, doesn't improve within the re-treatment period OR requires systemic treatment
  * Grade 3 drug-related uveitis, episcleritis, iritis, pneumonitis, bronchospasm, or neurologic toxicity
Time Frame: From first dose of study medication through 60 days following last dose of study treatment (assessed for an average of 7 months up to a max of approximately 27 months)
Population: All DLT Evaluable Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: BMS-986218 2 mg All Solid Tumors | Part 1A: BMS-986218 4 mg All Solid Tumors | Part 1A: BMS-986218 7 mg All Solid Tumors | Part 1A: BMS-986218 20 mg All Solid Tumors | Part 1A: BMS-986218 40 mg All Solid Tumors | Part 1A: BMS-986218 70 mg All Solid Tumors | Part 1A: BMS-986218 100 mg All Solid Tumors | Part 1A: BMS-986218 150 mg All Solid Tumors | Part 1A: BMS-986218 200 mg All Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors | Part 1A: BMS-986218 35 mg Select Solid Tumors | Part 1A: BMS-986218 50 mg Select Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors Pharmacodynamics Cohort | Part 1B: BMS-986218 7 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 20 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 40 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 70 mg + Nivolumab 480 mg Select Solid Tumors | Part 2A: Ipilimumab Cutaneous Melanoma | Part 2A: BMS-986218 7 mg Cutaneous Melanoma | Part 2A: BMS-986218 20 mg Cutaneous Melanoma | Part 2A: BMS-986218 70 mg Cutaneous Melanoma | Part 2B: BMS-986218 7 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 20 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 70 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2C: BMS-986218 + Nivolumab Non-Small Cell Lung Cancer (NSCLC) | Part 2D: BMS-986218 + Nivolumab Microsatellite Stable Colorectal Cancer (MSS CRC)
Number analyzed (Participants) | 4 | 9 | 11 | 13 | 10 | 12 | 7 | 11 | 5 | 14 | 5 | 4 | 1 | 5 | 14 | 16 | 7 | 3 | 3 | 2 | 2 | 6 | 7 | 4 | 18 | 18
Participants | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Adverse Events (AEs) Leading to Discontinuation
Description: as for outcome 1
Time Frame: as for outcome 1
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: BMS-986218 2 mg All Solid Tumors | Part 1A: BMS-986218 4 mg All Solid Tumors | Part 1A: BMS-986218 7 mg All Solid Tumors | Part 1A: BMS-986218 20 mg All Solid Tumors | Part 1A: BMS-986218 40 mg All Solid Tumors | Part 1A: BMS-986218 70 mg All Solid Tumors | Part 1A: BMS-986218 100 mg All Solid Tumors | Part 1A: BMS-986218 150 mg All Solid Tumors | Part 1A: BMS-986218 200 mg All Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors | Part 1A: BMS-986218 35 mg Select Solid Tumors | Part 1A: BMS-986218 50 mg Select Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors Pharmacodynamics Cohort | Part 1B: BMS-986218 7 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 20 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 40 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 70 mg + Nivolumab 480 mg Select Solid Tumors | Part 2A: Ipilimumab Cutaneous Melanoma | Part 2A: BMS-986218 7 mg Cutaneous Melanoma | Part 2A: BMS-986218 20 mg Cutaneous Melanoma | Part 2A: BMS-986218 70 mg Cutaneous Melanoma | Part 2B: BMS-986218 7 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 20 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 70 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2C: BMS-986218 + Nivolumab Non-Small Cell Lung Cancer (NSCLC) | Part 2D: BMS-986218 + Nivolumab Microsatellite Stable Colorectal Cancer (MSS CRC)
Number analyzed (Participants) | 4 | 9 | 12 | 15 | 12 | 14 | 7 | 11 | 5 | 14 | 6 | 4 | 1 | 5 | 17 | 19 | 7 | 20 | 19 | 18 | 18 | 22 | 22 | 22 | 29 | 44
Participants | 1 | 0 | 1 | 2 | 0 | 3 | 1 | 1 | 3 | 2 | 0 | 2 | 0 | 0 | 2 | 3 | 3 | 3 | 1 | 2 | 2 | 0 | 2 | 6 | 7 | 6

5. Primary Outcome: Number of Participants Who Died
Description: Number of participants who died during the study
Time Frame: From randomization (Part 2A and 2B) or first dose (Part 1, 2C and 2D) until study closure (Up to approximately 83 months)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: BMS-986218 2 mg All Solid Tumors | Part 1A: BMS-986218 4 mg All Solid Tumors | Part 1A: BMS-986218 7 mg All Solid Tumors | Part 1A: BMS-986218 20 mg All Solid Tumors | Part 1A: BMS-986218 40 mg All Solid Tumors | Part 1A: BMS-986218 70 mg All Solid Tumors | Part 1A: BMS-986218 100 mg All Solid Tumors | Part 1A: BMS-986218 150 mg All Solid Tumors | Part 1A: BMS-986218 200 mg All Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors | Part 1A: BMS-986218 35 mg Select Solid Tumors | Part 1A: BMS-986218 50 mg Select Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors Pharmacodynamics Cohort | Part 1B: BMS-986218 7 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 20 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 40 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 70 mg + Nivolumab 480 mg Select Solid Tumors | Part 2A: Ipilimumab Cutaneous Melanoma | Part 2A: BMS-986218 7 mg Cutaneous Melanoma | Part 2A: BMS-986218 20 mg Cutaneous Melanoma | Part 2A: BMS-986218 70 mg Cutaneous Melanoma | Part 2B: BMS-986218 7 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 20 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 70 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2C: BMS-986218 + Nivolumab Non-Small Cell Lung Cancer (NSCLC) | Part 2D: BMS-986218 + Nivolumab Microsatellite Stable Colorectal Cancer (MSS CRC)
Number analyzed (Participants) | 4 | 9 | 12 | 15 | 12 | 14 | 7 | 11 | 5 | 14 | 6 | 4 | 1 | 5 | 17 | 19 | 7 | 20 | 19 | 18 | 18 | 22 | 22 | 22 | 29 | 44
Participants | 2 | 7 | 6 | 10 | 8 | 7 | 6 | 10 | 1 | 9 | 6 | 3 | 1 | 4 | 15 | 14 | 5 | 13 | 16 | 16 | 18 | 19 | 20 | 16 | 28 | 37

6. Primary Outcome: Objective Response Rate (ORR) for Part 2 Only
Description: Objective response rate (ORR) is defined as the percent of all treated participants whose best overall response (BOR) is either complete response (CR) or partial response (PR) by Investigator per Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm (Note: The appearance of 1or more new lesions is also considered progression).
Time Frame: From the start of the study treatment until disease progression, or the last response recorded, taking into account any requirement for confirmation and censoring rules regarding subsequent therapy (Up to approximately 83 months)
Population: All Treated Participants
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Part 2A: Ipilimumab Cutaneous Melanoma | Part 2A: BMS-986218 7 mg Cutaneous Melanoma | Part 2A: BMS-986218 20 mg Cutaneous Melanoma | Part 2A: BMS-986218 70 mg Cutaneous Melanoma | Part 2B: BMS-986218 7 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 20 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 70 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2C: BMS-986218 + Nivolumab Non-Small Cell Lung Cancer (NSCLC) | Part 2D: BMS-986218 + Nivolumab Microsatellite Stable Colorectal Cancer (MSS CRC)
Number analyzed (Participants) | 20 | 19 | 18 | 18 | 22 | 22 | 22 | 29 | 44
Percent of participants | 25.0 [8.7 to 49.1] | 10.5 [1.3 to 33.1] | 5.6 [0.1 to 27.3] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 15.4] | 4.5 [0.1 to 22.8] | 4.5 [0.1 to 22.8] | 0.0 [0.0 to 11.9] | 4.5 [0.6 to 15.5]

7. Primary Outcome: Median Duration of Response (mDOR) for Part 2 Only
Description: Duration of response (DOR) for a participant with a BOR of CR or PR is defined as the time between the date of first response and the date of the first objectively documented tumor progression per RECIST v1.1 or death, whichever occurs first.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition, the sum must also demonstrate an absolute increase of at least 5mm (Note: The appearance of 1or more new lesions is also considered progression).
  Based on Kaplan-Meier estimates of duration of response
Time Frame: From the date of first dose to the date of the first objectively documented tumor progression, or death, whichever occurs first (Up to approximately 83 months)
Population: All confirmed responders in Part 2 whose best overall response (BOR) is either complete response (CR) or partial response (PR). Pre-specified to be reported for Part 2 only
Measure: Median (Full Range); unit: Months
Arm/Group | Part 2A: Ipilimumab Cutaneous Melanoma | Part 2A: BMS-986218 7 mg Cutaneous Melanoma | Part 2A: BMS-986218 20 mg Cutaneous Melanoma | Part 2A: BMS-986218 70 mg Cutaneous Melanoma | Part 2B: BMS-986218 7 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 20 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 70 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2C: BMS-986218 + Nivolumab Non-Small Cell Lung Cancer (NSCLC) | Part 2D: BMS-986218 + Nivolumab Microsatellite Stable Colorectal Cancer (MSS CRC)
Number analyzed (Participants) | 5 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 2
Months | 20.53 [3.65 to 20.53] | 4.75 [3.71 to 5.78] | 7.89 [7.89 to 7.89] |  |  | 5.52 [5.52 to 5.52] | NA [14.88 to 14.88] — Insufficient number of participants to calculate mDOR. Minimum and Maximum value was censored at the time of analysis. |  | NA [0.03 to 14.85] — Insufficient number of participants to calculate mDOR. Minimum and Maximum value was censored at the time of analysis.

8. Primary Outcome: Progression-free Survival Rate (PFSR) at 24, 36, and 48 Weeks for Part 2 Only
Description: Progression-free survival (PFS) for a participant is defined as the time from the first dosing date to the date of first objectively documented disease progression or death due to any cause, whichever occurs first.
  Based on Kaplan-Meier estimates of progression-free survival rate
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm (Note: The appearance of 1or more new lesions is also considered progression).
Time Frame: At 24, 36, and 48 weeks
Population: All treated participants for Part 2 only. Pre-specified to be reported for Part 2 only.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Part 2A: Ipilimumab Cutaneous Melanoma | Part 2A: BMS-986218 7 mg Cutaneous Melanoma | Part 2A: BMS-986218 20 mg Cutaneous Melanoma | Part 2A: BMS-986218 70 mg Cutaneous Melanoma | Part 2B: BMS-986218 7 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 20 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 70 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2C: BMS-986218 + Nivolumab Non-Small Cell Lung Cancer (NSCLC) | Part 2D: BMS-986218 + Nivolumab Microsatellite Stable Colorectal Cancer (MSS CRC)
Number analyzed (Participants) | 20 | 19 | 18 | 18 | 22 | 22 | 22 | 29 | 44
Percent of participants
  24 Weeks | 31.9 [13.1 to 52.6] | 22.2 [6.9 to 42.9] | 11.1 [1.9 to 29.8] | 11.1 [1.9 to 29.8] | 9.1 [1.6 to 25.1] | 16.3 [4.2 to 35.5] | 37.5 [15.8 to 59.4] | 11.7 [3.0 to 27] | 7.9 [2.0 to 19.0]
  36 Weeks | 19.1 [5.1 to 39.9] | 11.1 [1.9 to 29.8] | 11.1 [1.9 to 29.8] | 5.6 [0.4 to 22.4] | 9.1 [1.6 to 25.1] | 16.3 [4.2 to 35.5] | 18.8 [4.7 to 40.1] | 7.8 [1.4 to 22.0] | 7.9 [2.0 to 19.0]
  48 Weeks | 19.1 [5.1 to 39.9] | 5.6 [0.4 to 22.4] | 5.6 [0.4 to 22.4] | 5.6 [0.4 to 22.4] | 9.1 [1.6 to 25.1] | 5.4 [0.4 to 21.9] | 18.8 [4.7 to 40.1] | 7.8 [1.4 to 22.0] | 5.2 [1.0 to 15.4]

9. Secondary Outcome: Objective Response Rate (ORR) for Part1A and Part1B Only
Description: Objective response rate (ORR) is defined as the percent of all treated participants whose best overall response (BOR) is either complete response (CR) or partial response (PR) by Investigator per Response Evaluation Criteria in Solid Tumors (RECIST v1.1)
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm (Note: The appearance of 1or more new lesions is also considered progression).
Time Frame: as for outcome 6
Population: All treated participants in Part1A and Part1B. Pre-specified to be collected for Part1A and Part1B only.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Part 1A: BMS-986218 2 mg All Solid Tumors | Part 1A: BMS-986218 4 mg All Solid Tumors | Part 1A: BMS-986218 7 mg All Solid Tumors | Part 1A: BMS-986218 20 mg All Solid Tumors | Part 1A: BMS-986218 40 mg All Solid Tumors | Part 1A: BMS-986218 70 mg All Solid Tumors | Part 1A: BMS-986218 100 mg All Solid Tumors | Part 1A: BMS-986218 150 mg All Solid Tumors | Part 1A: BMS-986218 200 mg All Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors | Part 1A: BMS-986218 35 mg Select Solid Tumors | Part 1A: BMS-986218 50 mg Select Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors Pharmacodynamics Cohort | Part 1B: BMS-986218 7 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 20 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 40 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 70 mg + Nivolumab 480 mg Select Solid Tumors
Number analyzed (Participants) | 4 | 9 | 12 | 15 | 12 | 14 | 7 | 11 | 5 | 14 | 6 | 4 | 1 | 5 | 17 | 19 | 7
Percent of participants | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 23.2] | 14.3 [0.4 to 57.9] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 52.2] | 7.1 [0.2 to 33.9] | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 52.2] | 0.0 [0.0 to 19.5] | 5.3 [0.1 to 26.0] | 28.6 [3.7 to 71.0]

10. Secondary Outcome: Median Duration of Response (mDOR) for Part1A and Part1B Only
Description: as for outcome 7
Time Frame: as for outcome 7
Population: All treated participants in Part1A and Part1B. Pre-specified to be collected for Part1A and Part1B only.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Part 1A: BMS-986218 2 mg All Solid Tumors | Part 1A: BMS-986218 4 mg All Solid Tumors | Part 1A: BMS-986218 7 mg All Solid Tumors | Part 1A: BMS-986218 20 mg All Solid Tumors | Part 1A: BMS-986218 40 mg All Solid Tumors | Part 1A: BMS-986218 70 mg All Solid Tumors | Part 1A: BMS-986218 100 mg All Solid Tumors | Part 1A: BMS-986218 150 mg All Solid Tumors | Part 1A: BMS-986218 200 mg All Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors | Part 1A: BMS-986218 35 mg Select Solid Tumors | Part 1A: BMS-986218 50 mg Select Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors Pharmacodynamics Cohort | Part 1B: BMS-986218 7 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 20 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 40 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 70 mg + Nivolumab 480 mg Select Solid Tumors
Number analyzed (Participants) | 4 | 9 | 12 | 15 | 12 | 14 | 7 | 11 | 5 | 14 | 6 | 4 | 1 | 5 | 17 | 19 | 7
Percent of participants | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 23.2] | 14.3 [0.4 to 57.9] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 52.2] | 7.1 [0.2 to 33.9] | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 52.2] | 0.0 [0.0 to 19.5] | 5.3 [0.1 to 26.0] | 28.6 [3.7 to 71.0]

11. Secondary Outcome: Progression-free Survival Rate (PFSR) at 24, 36, and 48 Weeks for Part1A and Part1B Only
Description: Progression-free survival (PFS) for a participant is defined as the time from the first dosing date to the date of first objectively documented disease progression or death due to any cause, whichever occurs first.
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition, the sum must also demonstrate an absolute increase of at least 5mm (Note: The appearance of 1or more new lesions is also considered progression).
  Based on Kaplan-Meier estimates of progression-free survival rate
Time Frame: At 24, 36, and 48 weeks
Population: All treated participants in Part1A and Part1B. Pre-specified to be collected for Part1A and Part1B only.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Part 1A: BMS-986218 2 mg All Solid Tumors | Part 1A: BMS-986218 4 mg All Solid Tumors | Part 1A: BMS-986218 7 mg All Solid Tumors | Part 1A: BMS-986218 20 mg All Solid Tumors | Part 1A: BMS-986218 40 mg All Solid Tumors | Part 1A: BMS-986218 70 mg All Solid Tumors | Part 1A: BMS-986218 100 mg All Solid Tumors | Part 1A: BMS-986218 150 mg All Solid Tumors | Part 1A: BMS-986218 200 mg All Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors | Part 1A: BMS-986218 35 mg Select Solid Tumors | Part 1A: BMS-986218 50 mg Select Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors Pharmacodynamics Cohort | Part 1B: BMS-986218 7 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 20 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 40 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 70 mg + Nivolumab 480 mg Select Solid Tumors
Number analyzed (Participants) | 4 | 9 | 12 | 15 | 12 | 14 | 7 | 11 | 5 | 14 | 6 | 4 | 1 | 5 | 17 | 19 | 7
Percent of participants
  24 Weeks | 33.3 [0.9 to 77.4] | 22.2 [3.4 to 51.3] | 16.7 [2.7 to 41.3] | 15.4 [2.5 to 38.8] | 9.1 [0.5 to 33.3] | 0.0 [0.0 to 0.0] | 17.1 [0.8 to 52.6] | 9.1 [0.5 to 33.3] | 0.0 [0.0 to 0.0] | 7.1 [0.5 to 27.5] | 16.7 [0.8 to 51.7] | 50.0 [5.8 to 84.5] | 0.0 [0.0 to 0.0] | 20.0 [0.8 to 58.2] | 9.5 [0.6 to 33.5] | 11.1 [1.9 to 29.8] | 28.6 [4.1 to 61.2]
  36 Weeks: number analyzed (Participants) | 4 | 9 | 12 | 15 | 12 | 14 | 0 | 11 | 5 | 14 | 6 | 4 | 1 | 5 | 17 | 19 | 7
  36 Weeks | 0.0 [0.0 to 0.0] | 22.2 [3.4 to 51.3] | 0.0 [0.0 to 0.0] | 7.7 [0.5 to 29.2] | 9.1 [0.5 to 33.3] | 0.0 [0.0 to 0.0] |  | 9.1 [0.5 to 33.3] | 0.0 [0.0 to 0.0] | 7.1 [0.5 to 27.5] | 0.0 [0.0 to 0.0] | 50.0 [5.8 to 84.5] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 11.1 [1.9 to 29.8] | 28.6 [4.1 to 61.2]
  48 Weeks: number analyzed (Participants) | 4 | 9 | 12 | 15 | 12 | 14 | 0 | 11 | 5 | 14 | 6 | 4 | 1 | 5 | 17 | 19 | 7
  48 Weeks | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 7.7 [0.5 to 29.2] | 9.1 [0.5 to 33.3] | 0.0 [0.0 to 0.0] |  | 9.1 [0.5 to 33.3] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 11.1 [1.9 to 29.8] | 28.6 [4.1 to 61.2]

12. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) for BMS-986218
Description: Cmax is the maximum observed serum concentration for BMS-986218.
Time Frame: On Cycle 1 Day 1, Cycle 1 Day 15, Cycle 3 Day 1, Cycle 3 Day 15 (Each Cycle is of 28 Days)
Population: All PK participants with available BMS-986218 PK results at each time point. Participants in Part 2A Ipilimumab Cutaneous Melanoma did not receive BMS-986218 and hence BMS-986218 PK data can not be reported for this group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1A: BMS-986218 2 mg All Solid Tumors | Part 1A: BMS-986218 4 mg All Solid Tumors | Part 1A: BMS-986218 7 mg All Solid Tumors | Part 1A: BMS-986218 20 mg All Solid Tumors | Part 1A: BMS-986218 40 mg All Solid Tumors | Part 1A: BMS-986218 70 mg All Solid Tumors | Part 1A: BMS-986218 100 mg All Solid Tumors | Part 1A: BMS-986218 150 mg All Solid Tumors | Part 1A: BMS-986218 200 mg All Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors | Part 1A: BMS-986218 35 mg Select Solid Tumors | Part 1A: BMS-986218 50 mg Select Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors Pharmacodynamics Cohort | Part 1B: BMS-986218 7 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 20 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 40 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 70 mg + Nivolumab 480 mg Select Solid Tumors | Part 2A: Ipilimumab Cutaneous Melanoma | Part 2A: BMS-986218 7 mg Cutaneous Melanoma | Part 2A: BMS-986218 20 mg Cutaneous Melanoma | Part 2A: BMS-986218 70 mg Cutaneous Melanoma | Part 2B: BMS-986218 7 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 20 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 70 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2C: BMS-986218 + Nivolumab Non-Small Cell Lung Cancer (NSCLC) | Part 2D: BMS-986218 + Nivolumab Microsatellite Stable Colorectal Cancer (MSS CRC)
Number analyzed (Participants) | 4 | 9 | 12 | 15 | 12 | 14 | 7 | 11 | 5 | 14 | 6 | 4 | 1 | 5 | 17 | 18 | 7 | 0 | 15 | 17 | 17 | 20 | 20 | 20 | 27 | 41
ng/mL
  Cycle 1 Day 1 | 378.20 (69.94) | 898.37 (35.77) | 1918.89 (27.17) | 5162.91 (31.89) | 10167.06 (34.47) | 19191.31 (23.63) | 28404.67 (25.91) | 38955.95 (46.84) | 34268.86 (30.14) | 5198.38 (23.13) | 6774.51 (32.40) | 13852.30 (22.40) | 3800.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 2196.42 (34.99) | 4009.69 (40.55) | 7672.60 (39.22) | 17399.93 (29.04) |  | 2096.56 (42.66) | 4759.66 (46.15) | 17121.28 (22.99) | 2207.18 (102.83) | 5890.68 (60.79) | 16114.18 (37.86) | 9545.23 (39.78) | 8977.53 (38.23)
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 15 |  |  |  |  |  |  |  |  |  | 6039.57 (32.03) | 8958.71 (30.62) | 17041.16 (16.18) |  |  |  |  |  |  |  |  |  |  |  |  |  |
  Cycle 3 Day 1: number analyzed (Participants) | 2 | 4 | 6 | 4 | 4 | 2 | 3 | 4 | 0 | 3 | 2 | 2 | 1 | 2 | 4 | 7 | 1 | 0 | 13 | 12 | 8 | 11 | 12 | 10 | 11 | 9
  Cycle 3 Day 1 | 636.63 (12.17) | 1041.61 (22.08) | 1984.34 (20.51) | 5013.30 (40.59) | 9461.39 (51.18) | 23878.44 (10.92) | 26728.01 (38.43) | 40591.79 (11.96) |  | 5198.25 (15.55) | 9896.67 (9.69) | 17526.84 (32.21) | 5870.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 1849.00 (25.58) | 3568.33 (47.96) | 7900.78 (29.53) | 14300.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation |  | 2430.88 (30.45) | 7837.32 (169.78) | 16491.17 (26.01) | 2812.74 (52.12) | 6236.74 (37.92) | 23527.72 (50.87) | 10711.87 (28.93) | 10317.85 (42.91)
  Cycle 3 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 3 Day 15 |  |  |  |  |  |  |  |  |  | 5485.98 (30.70) | 9090.35 (13.17) | 13100.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 6540.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation |  |  |  |  |  |  |  |  |  |  |  |  |

13. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration [AUC(0-T)] for BMS-986218
Description: Tmax is the time taken to reach the maximum observed serum concentration (Cmax) for BMS-986218.
Time Frame: On Cycle 1 Day 1, Cycle 1 Day 15, Cycle 3 Day 1, Cycle 3 Day 15 (Each Cycle is of 28 Days)
Population: All PK participants with available PK results at each time point
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1A: BMS-986218 2 mg All Solid Tumors | Part 1A: BMS-986218 4 mg All Solid Tumors | Part 1A: BMS-986218 7 mg All Solid Tumors | Part 1A: BMS-986218 20 mg All Solid Tumors | Part 1A: BMS-986218 40 mg All Solid Tumors | Part 1A: BMS-986218 70 mg All Solid Tumors | Part 1A: BMS-986218 100 mg All Solid Tumors | Part 1A: BMS-986218 150 mg All Solid Tumors | Part 1A: BMS-986218 200 mg All Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors | Part 1A: BMS-986218 35 mg Select Solid Tumors | Part 1A: BMS-986218 50 mg Select Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors Pharmacodynamics Cohort | Part 1B: BMS-986218 7 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 20 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 40 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 70 mg + Nivolumab 480 mg Select Solid Tumors | Part 2A: Ipilimumab Cutaneous Melanoma | Part 2A: BMS-986218 7 mg Cutaneous Melanoma | Part 2A: BMS-986218 20 mg Cutaneous Melanoma | Part 2A: BMS-986218 70 mg Cutaneous Melanoma | Part 2B: BMS-986218 7 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 20 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 70 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2C: BMS-986218 + Nivolumab Non-Small Cell Lung Cancer (NSCLC) | Part 2D: BMS-986218 + Nivolumab Microsatellite Stable Colorectal Cancer (MSS CRC)
Number analyzed (Participants) | 4 | 9 | 12 | 15 | 12 | 14 | 7 | 11 | 5 | 14 | 6 | 4 | 1 | 5 | 17 | 18 | 7 | 0 | 15 | 17 | 17 | 20 | 20 | 20 | 27 | 41
h*ng/mL
  Cycle 1 Day 1 | 38482.79 (67.05) | 152995.20 (24.90) | 338090.13 (44.06) | 859624.01 (35.00) | 1374751.12 (41.91) | 2800743.92 (34.47) | 4813781.16 (28.58) | 6332567.97 (32.76) | 6471486.44 (42.01) | 555237.58 (35.05) | 911929.11 (36.66) | 1878893.05 (27.29) | 698634.55 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 346844.14 (43.83) | 568755.53 (50.38) | 1196906.59 (39.01) | 2675458.62 (25.81) |  | 362116.78 (42.58) | 1001283.21 (50.58) | 3086017.57 (21.62) | 352268.83 (78.80) | 1067646.86 (40.62) | 2733292.53 (35.02) | 1461119.11 (35.96) | 1380362.22 (42.32)
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 15 |  |  |  |  |  |  |  |  |  | 666441.31 (50.63) | 812419.15 (67.75) | 2710445.36 (7.15) |  |  |  |  |  |  |  |  |  |  |  |  |  |
  Cycle 3 Day 1: number analyzed (Participants) | 2 | 4 | 6 | 4 | 4 | 2 | 3 | 4 | 0 | 3 | 2 | 2 | 1 | 2 | 4 | 7 | 1 | 0 | 13 | 12 | 8 | 11 | 12 | 10 | 11 | 9
  Cycle 3 Day 1 | 106995.38 (25.94) | 180870.63 (13.77) | 320865.91 (52.33) | 916409.73 (31.83) | 1231569.13 (60.51) | 4712195.98 (22.69) | 4496192.21 (30.37) | 7327105.74 (35.84) |  | 829253.53 (24.59) | 1673664.31 (29.67) | 1162456.20 (123.44) | 1058967.60 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 284245.76 (46.27) | 586413.48 (57.48) | 1530718.58 (31.46) | 2090995.50 (NA) — Insufficient number of participants to calculate geometric coefficient of variation |  | 242498.24 (71.75) | 1070790.34 (205.76) | 2152498.70 (42.12) | 303622.32 (52.88) | 982950.43 (51.34) | 3653192.45 (34.54) | 1609530.93 (45.25) | 1716552.20 (22.69)
  Cycle 3 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 3 Day 15 |  |  |  |  |  |  |  |  |  | 753989.60 (57.54) | 1853267.79 (11.48) | 1619652.01 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 732535.33 (NA) — Insufficient number of participants to calculate geometric coefficient of variation |  |  |  |  |  |  |  |  |  |  |  |  |

14. Secondary Outcome: Area Under the Concentration-time Curve in 1 Dosing Interval [AUC(TAU)] for BMS-986218
Description: AUC (TAU) is the area measured under the concentration-time curve taken over the dosing interval for BMS-986218.
Time Frame: On Cycle 1 Day 1, Cycle 1 Day 15, Cycle 3 Day 1, Cycle 3 Day 15 (Each Cycle is of 28 Days)
Population: All PK participants with available PK results at each time point
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1A: BMS-986218 2 mg All Solid Tumors | Part 1A: BMS-986218 4 mg All Solid Tumors | Part 1A: BMS-986218 7 mg All Solid Tumors | Part 1A: BMS-986218 20 mg All Solid Tumors | Part 1A: BMS-986218 40 mg All Solid Tumors | Part 1A: BMS-986218 70 mg All Solid Tumors | Part 1A: BMS-986218 100 mg All Solid Tumors | Part 1A: BMS-986218 150 mg All Solid Tumors | Part 1A: BMS-986218 200 mg All Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors | Part 1A: BMS-986218 35 mg Select Solid Tumors | Part 1A: BMS-986218 50 mg Select Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors Pharmacodynamics Cohort | Part 1B: BMS-986218 7 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 20 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 40 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 70 mg + Nivolumab 480 mg Select Solid Tumors | Part 2A: Ipilimumab Cutaneous Melanoma | Part 2A: BMS-986218 7 mg Cutaneous Melanoma | Part 2A: BMS-986218 20 mg Cutaneous Melanoma | Part 2A: BMS-986218 70 mg Cutaneous Melanoma | Part 2B: BMS-986218 7 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 20 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 70 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2C: BMS-986218 + Nivolumab Non-Small Cell Lung Cancer (NSCLC) | Part 2D: BMS-986218 + Nivolumab Microsatellite Stable Colorectal Cancer (MSS CRC)
Number analyzed (Participants) | 2 | 9 | 11 | 13 | 11 | 14 | 7 | 10 | 4 | 11 | 5 | 4 | 1 | 5 | 14 | 15 | 7 | 0 | 15 | 16 | 17 | 20 | 20 | 19 | 26 | 36
h*ng/mL
  Cycle 1 Day 1 | 102107.56 (20.44) | 160708.57 (21.45) | 376035.72 (38.14) | 894413.40 (35.17) | 1421515.99 (40.74) | 3027482.69 (33.30) | 4816815.14 (23.87) | 6599896.79 (22.75) | 7560614.03 (28.48) | 604538.01 (32.38) | 984127.10 (33.75) | 1878893.05 (27.29) | 698634.55 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 346844.14 (43.83) | 765535.55 (37.86) | 1400907.18 (31.92) | 2736051.44 (25.50) |  | 355092.73 (43.60) | 1107418.00 (43.18) | 3074048.83 (19.62) | 366958.19 (75.83) | 1096040.02 (38.84) | 2884299.15 (30.80) | 1488804.73 (35.18) | 1516016.83 (38.72)
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 15 |  |  |  |  |  |  |  |  |  | 791252.01 (42.41) | 1254494.19 (41.07) | 2710445.36 (7.15) |  |  |  |  |  |  |  |  |  |  |  |  |  |
  Cycle 3 Day 1: number analyzed (Participants) | 2 | 4 | 5 | 3 | 4 | 1 | 2 | 4 | 0 | 3 | 2 | 1 | 1 | 2 | 3 | 6 | 1 | 0 | 10 | 8 | 6 | 7 | 10 | 10 | 11 | 9
  Cycle 3 Day 1 | 110809.32 (21.12) | 189406.70 (12.74) | 460618.56 (29.45) | 946000.30 (44.09) | 1265811.65 (67.93) | 4008112.03 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 5131052.16 (1.63) | 7635138.59 (31.66) |  | 829253.53 (24.59) | 1673664.31 (29.67) | 3363278.02 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 1058967.60 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 284245.76 (46.27) | 827831.27 (33.07) | 1569751.67 (32.78) | 2090995.50 (NA) — Insufficient number of participants to calculate geometric coefficient of variation |  | 438160.20 (44.33) | 1777132.02 (156.77) | 2986930.70 (24.50) | 471293.82 (33.36) | 1189672.74 (38.19) | 3636946.89 (34.65) | 1650434.22 (44.45) | 1760069.89 (26.26)
  Cycle 3 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 3 Day 15 |  |  |  |  |  |  |  |  |  | 1161185.91 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 1853267.79 (11.48) |  |  |  |  |  |  |  |  |  |  |  |  |  |  |

15. Secondary Outcome: Observed Concentration at the End of a Dosing Interval (Ctau) for BMS-986218
Description: Ctau is the observed serum concentration at the end of the dosing interval for BMS-986218.
Time Frame: On Cycle 1 Day 1, Cycle 1 Day 15, Cycle 3 Day 1, Cycle 3 Day 15 (Each Cycle is of 28 Days)
Population: All PK participants with available PK results at each time point
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1A: BMS-986218 2 mg All Solid Tumors | Part 1A: BMS-986218 4 mg All Solid Tumors | Part 1A: BMS-986218 7 mg All Solid Tumors | Part 1A: BMS-986218 20 mg All Solid Tumors | Part 1A: BMS-986218 40 mg All Solid Tumors | Part 1A: BMS-986218 70 mg All Solid Tumors | Part 1A: BMS-986218 100 mg All Solid Tumors | Part 1A: BMS-986218 150 mg All Solid Tumors | Part 1A: BMS-986218 200 mg All Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors | Part 1A: BMS-986218 35 mg Select Solid Tumors | Part 1A: BMS-986218 50 mg Select Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors Pharmacodynamics Cohort | Part 1B: BMS-986218 7 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 20 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 40 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 70 mg + Nivolumab 480 mg Select Solid Tumors | Part 2A: Ipilimumab Cutaneous Melanoma | Part 2A: BMS-986218 7 mg Cutaneous Melanoma | Part 2A: BMS-986218 20 mg Cutaneous Melanoma | Part 2A: BMS-986218 70 mg Cutaneous Melanoma | Part 2B: BMS-986218 7 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 20 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 70 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2C: BMS-986218 + Nivolumab Non-Small Cell Lung Cancer (NSCLC) | Part 2D: BMS-986218 + Nivolumab Microsatellite Stable Colorectal Cancer (MSS CRC)
Number analyzed (Participants) | 2 | 9 | 11 | 13 | 11 | 14 | 7 | 10 | 4 | 11 | 5 | 4 | 1 | 5 | 14 | 15 | 7 | 0 | 15 | 16 | 17 | 20 | 20 | 19 | 26 | 36
ng/mL
  Cycle 1 Day 1 | 39.29 (18.84) | 54.25 (46.26) | 184.40 (53.72) | 304.84 (66.34) | 293.28 (82.69) | 792.03 (76.23) | 1600.37 (31.94) | 2396.65 (51.08) | 2659.87 (32.41) | 703.99 (45.94) | 1284.78 (42.93) | 2793.34 (31.31) | 1090.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 99.96 (45.22) | 176.14 (63.80) | 466.01 (67.94) | 667.59 (62.14) |  | 140.54 (62.61) | 530.35 (144.43) | 959.00 (56.06) | 133.30 (118.13) | 379.50 (62.15) | 810.78 (69.02) | 330.53 (65.42) | 341.97 (74.43)
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 15 |  |  |  |  |  |  |  |  |  | 1016.63 (57.51) | 1651.22 (51.66) | 3630.54 (21.56) |  |  |  |  |  |  |  |  |  |  |  |  |  |
  Cycle 3 Day 1: number analyzed (Participants) | 2 | 4 | 5 | 3 | 4 | 1 | 2 | 4 | 0 | 3 | 2 | 1 | 1 | 2 | 3 | 6 | 1 | 0 | 10 | 8 | 6 | 7 | 10 | 10 | 11 | 9
  Cycle 3 Day 1 | 43.06 (73.10) | 88.58 (30.12) | 239.24 (37.53) | 275.23 (54.82) | 262.71 (106.82) | 2310.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 2089.02 (33.02) | 3151.12 (64.09) |  | 1098.35 (31.92) | 2723.07 (23.06) | 5161.39 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 1550.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 140.76 (67.67) | 294.67 (34.83) | 559.93 (63.00) | 339.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation |  | 154.17 (76.15) | 795.20 (166.56) | 1033.06 (33.10) | 195.37 (39.51) | 442.46 (66.32) | 1326.75 (50.09) | 423.20 (85.57) | 516.44 (58.12)
  Cycle 3 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 3 Day 15 |  |  |  |  |  |  |  |  |  | 1980.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 3212.85 (27.42) |  |  |  |  |  |  |  |  |  |  |  |  |  |  |

16. Secondary Outcome: Total Body Clearance (CLT/F) for BMS-986218
Time Frame: At Cycle 3 Day 1 (Each Cycle is of 28 Days)
Population: All treated participants with total body clearance were measured at Cycle 3 Day 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h
Arm/Group | Part 1A: BMS-986218 2 mg All Solid Tumors | Part 1A: BMS-986218 4 mg All Solid Tumors | Part 1A: BMS-986218 7 mg All Solid Tumors | Part 1A: BMS-986218 20 mg All Solid Tumors | Part 1A: BMS-986218 40 mg All Solid Tumors | Part 1A: BMS-986218 70 mg All Solid Tumors | Part 1A: BMS-986218 100 mg All Solid Tumors | Part 1A: BMS-986218 150 mg All Solid Tumors | Part 1A: BMS-986218 200 mg All Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors | Part 1A: BMS-986218 35 mg Select Solid Tumors | Part 1A: BMS-986218 50 mg Select Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors Pharmacodynamics Cohort | Part 1B: BMS-986218 7 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 20 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 40 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 70 mg + Nivolumab 480 mg Select Solid Tumors | Part 2A: Ipilimumab Cutaneous Melanoma | Part 2A: BMS-986218 7 mg Cutaneous Melanoma | Part 2A: BMS-986218 20 mg Cutaneous Melanoma | Part 2A: BMS-986218 70 mg Cutaneous Melanoma | Part 2B: BMS-986218 7 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 20 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 70 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2C: BMS-986218 + Nivolumab Non-Small Cell Lung Cancer (NSCLC) | Part 2D: BMS-986218 + Nivolumab Microsatellite Stable Colorectal Cancer (MSS CRC)
Number analyzed (Participants) | 2 | 4 | 5 | 3 | 4 | 1 | 2 | 4 | 0 | 3 | 2 | 1 | 1 | 2 | 3 | 6 | 1 | 0 | 10 | 8 | 6 | 7 | 10 | 10 | 11 | 9
mL/h | 18.05 (21.12) | 21.12 (13.87) | 15.20 (43.36) | 21.14 (59.06) | 31.60 (61.89) | 17.46 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 19.49 (1.63) | 19.65 (30.54) |  | 24.12 (22.83) | 20.91 (29.67) | 14.87 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 18.89 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 24.63 (46.27) | 24.16 (40.86) | 25.48 (37.36) | 33.48 (NA) — Insufficient number of participants to calculate geometric coefficient of variation |  | 15.98 (51.15) | 11.25 (57.31) | 23.44 (31.87) | 14.85 (27.95) | 16.81 (33.59) | 19.25 (45.86) | 24.24 (60.65) | 22.73 (20.24)

17. Secondary Outcome: Average Concentration Over a Dosing Interval (AUC[TAU]/Tau) at Steady State (Css-avg) for BMS-986218
Time Frame: At Cycle 3 Day 1 (Each Cycle is of 28 Days)
Population: All treated participants with average concentration over a dosing interval at steady state were measured at Cycle 3 Day 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1A: BMS-986218 2 mg All Solid Tumors | Part 1A: BMS-986218 4 mg All Solid Tumors | Part 1A: BMS-986218 7 mg All Solid Tumors | Part 1A: BMS-986218 20 mg All Solid Tumors | Part 1A: BMS-986218 40 mg All Solid Tumors | Part 1A: BMS-986218 70 mg All Solid Tumors | Part 1A: BMS-986218 100 mg All Solid Tumors | Part 1A: BMS-986218 150 mg All Solid Tumors | Part 1A: BMS-986218 200 mg All Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors | Part 1A: BMS-986218 35 mg Select Solid Tumors | Part 1A: BMS-986218 50 mg Select Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors Pharmacodynamics Cohort | Part 1B: BMS-986218 7 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 20 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 40 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 70 mg + Nivolumab 480 mg Select Solid Tumors | Part 2A: Ipilimumab Cutaneous Melanoma | Part 2A: BMS-986218 7 mg Cutaneous Melanoma | Part 2A: BMS-986218 20 mg Cutaneous Melanoma | Part 2A: BMS-986218 70 mg Cutaneous Melanoma | Part 2B: BMS-986218 7 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 20 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 70 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2C: BMS-986218 + Nivolumab Non-Small Cell Lung Cancer (NSCLC) | Part 2D: BMS-986218 + Nivolumab Microsatellite Stable Colorectal Cancer (MSS CRC)
Number analyzed (Participants) | 2 | 4 | 5 | 3 | 4 | 1 | 2 | 4 | 0 | 3 | 2 | 1 | 1 | 2 | 3 | 6 | 1 | 0 | 10 | 8 | 6 | 7 | 10 | 10 | 11 | 9
ng/mL | 165.22 (21.39) | 282.04 (12.75) | 686.31 (29.48) | 1393.64 (45.15) | 1881.64 (68.23) | 5980.92 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 7644.60 (1.80) | 11589.37 (35.71) |  | 2420.43 (20.98) | 5006.22 (29.63) | 10009.76 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 3142.64 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 448.98 (43.83) | 1234.39 (32.97) | 2334.85 (32.57) | 2490.67 (NA) — Insufficient number of participants to calculate geometric coefficient of variation |  | 659.08 (44.76) | 2633.76 (157.01) | 4303.25 (21.87) | 685.48 (34.93) | 1760.14 (35.04) | 5347.42 (32.03) | 2429.04 (43.75) | 2627.53 (26.08)

18. Secondary Outcome: Ratio of an Exposure Measure at Steady State to That After the First Dose (Exposure Measure Includes Cmax) (AI_Cmax) for BMS-986218
Time Frame: At Cycle 3 Day 1 (Each Cycle is of 28 Days)
Population: All treated participants with ratio of an exposure measure at steady state to that after the first dose (exposure measure includes Cmax) were measured at Cycle 3 Day 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1A: BMS-986218 2 mg All Solid Tumors | Part 1A: BMS-986218 4 mg All Solid Tumors | Part 1A: BMS-986218 7 mg All Solid Tumors | Part 1A: BMS-986218 20 mg All Solid Tumors | Part 1A: BMS-986218 40 mg All Solid Tumors | Part 1A: BMS-986218 70 mg All Solid Tumors | Part 1A: BMS-986218 100 mg All Solid Tumors | Part 1A: BMS-986218 150 mg All Solid Tumors | Part 1A: BMS-986218 200 mg All Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors | Part 1A: BMS-986218 35 mg Select Solid Tumors | Part 1A: BMS-986218 50 mg Select Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors Pharmacodynamics Cohort | Part 1B: BMS-986218 7 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 20 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 40 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 70 mg + Nivolumab 480 mg Select Solid Tumors | Part 2A: Ipilimumab Cutaneous Melanoma | Part 2A: BMS-986218 7 mg Cutaneous Melanoma | Part 2A: BMS-986218 20 mg Cutaneous Melanoma | Part 2A: BMS-986218 70 mg Cutaneous Melanoma | Part 2B: BMS-986218 7 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 20 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 70 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2C: BMS-986218 + Nivolumab Non-Small Cell Lung Cancer (NSCLC) | Part 2D: BMS-986218 + Nivolumab Microsatellite Stable Colorectal Cancer (MSS CRC)
Number analyzed (Participants) | 2 | 4 | 6 | 4 | 4 | 2 | 3 | 4 | 0 | 3 | 2 | 2 | 1 | 2 | 4 | 7 | 1 | 0 | 12 | 12 | 8 | 10 | 12 | 10 | 11 | 9
Ratio | 0.83 (10.89) | 1.15 (22.83) | 1.13 (22.62) | 1.22 (52.14) | 0.91 (6.40) | 1.10 (8.26) | 0.77 (39.73) | 1.32 (1.53) |  | 1.12 (8.28) | 1.26 (53.95) | 1.29 (5.21) | 1.54 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 1.07 (8.70) | 0.77 (37.44) | 0.84 (27.10) | 1.08 (NA) — Insufficient number of participants to calculate geometric coefficient of variation |  | 1.19 (80.37) | 1.71 (115.10) | 0.90 (21.26) | 1.33 (93.11) | 1.00 (52.38) | 1.45 (136.48) | 1.05 (20.63) | 1.18 (40.84)

19. Secondary Outcome: Accumulation Index Ratio of AUC at Steady State to That After the First Dose (AI_AUC) for BMS-986218
Time Frame: At Cycle 3 Day 1 (Each Cycle is of 28 Days)
Population: All treated participants with accumulation index ratio of AUC at steady state to that after the first dose were measured at Cycle 3 Day 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1A: BMS-986218 2 mg All Solid Tumors | Part 1A: BMS-986218 4 mg All Solid Tumors | Part 1A: BMS-986218 7 mg All Solid Tumors | Part 1A: BMS-986218 20 mg All Solid Tumors | Part 1A: BMS-986218 40 mg All Solid Tumors | Part 1A: BMS-986218 70 mg All Solid Tumors | Part 1A: BMS-986218 100 mg All Solid Tumors | Part 1A: BMS-986218 150 mg All Solid Tumors | Part 1A: BMS-986218 200 mg All Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors | Part 1A: BMS-986218 35 mg Select Solid Tumors | Part 1A: BMS-986218 50 mg Select Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors Pharmacodynamics Cohort | Part 1B: BMS-986218 7 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 20 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 40 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 70 mg + Nivolumab 480 mg Select Solid Tumors | Part 2A: Ipilimumab Cutaneous Melanoma | Part 2A: BMS-986218 7 mg Cutaneous Melanoma | Part 2A: BMS-986218 20 mg Cutaneous Melanoma | Part 2A: BMS-986218 70 mg Cutaneous Melanoma | Part 2B: BMS-986218 7 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 20 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 70 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2C: BMS-986218 + Nivolumab Non-Small Cell Lung Cancer (NSCLC) | Part 2D: BMS-986218 + Nivolumab Microsatellite Stable Colorectal Cancer (MSS CRC)
Number analyzed (Participants) | 2 | 4 | 5 | 3 | 4 | 1 | 2 | 4 | 0 | 2 | 2 | 1 | 1 | 2 | 3 | 6 | 1 | 0 | 9 | 8 | 6 | 7 | 10 | 10 | 11 | 9
Ratio | 1.09 (0.69) | 1.16 (28.89) | 1.43 (26.71) | 1.29 (25.00) | 0.81 (17.94) | 1.16 (NA) — Insufficient number of participants to calculate Geometric mean and Geometric coefficient of variation | 1.09 (8.11) | 1.16 (17.02) |  | 1.49 (2.93) | 1.43 (54.87) | 1.28 (NA) — Insufficient number of participants to calculate Geometric mean and Geometric coefficient of variation | 1.52 (NA) — Insufficient number of participants to calculate Geometric mean and Geometric coefficient of variation | 1.09 (15.24) | 1.09 (15.52) | 1.13 (13.09) | 1.13 (NA) — Insufficient number of participants to calculate Geometric mean and Geometric coefficient of variation |  | 1.36 (96.87) | 1.37 (104.97) | 0.93 (25.69) | 1.48 (47.11) | 0.98 (34.75) | 1.29 (27.70) | 1.04 (19.75) | 1.18 (31.02)

20. Secondary Outcome: Terminal Serum Half-life (T-HALF) for BMS-986218
Time Frame: At Cycle 3 Day 1 (Each Cycle is of 28 Days)
Population: All treated participants with terminal serum half-life were measured at Cycle 3 Day 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Part 1A: BMS-986218 2 mg All Solid Tumors | Part 1A: BMS-986218 4 mg All Solid Tumors | Part 1A: BMS-986218 7 mg All Solid Tumors | Part 1A: BMS-986218 20 mg All Solid Tumors | Part 1A: BMS-986218 40 mg All Solid Tumors | Part 1A: BMS-986218 70 mg All Solid Tumors | Part 1A: BMS-986218 100 mg All Solid Tumors | Part 1A: BMS-986218 150 mg All Solid Tumors | Part 1A: BMS-986218 200 mg All Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors | Part 1A: BMS-986218 35 mg Select Solid Tumors | Part 1A: BMS-986218 50 mg Select Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors Pharmacodynamics Cohort | Part 1B: BMS-986218 7 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 20 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 40 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 70 mg + Nivolumab 480 mg Select Solid Tumors | Part 2A: Ipilimumab Cutaneous Melanoma | Part 2A: BMS-986218 7 mg Cutaneous Melanoma | Part 2A: BMS-986218 20 mg Cutaneous Melanoma | Part 2A: BMS-986218 70 mg Cutaneous Melanoma | Part 2B: BMS-986218 7 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 20 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 70 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2C: BMS-986218 + Nivolumab Non-Small Cell Lung Cancer (NSCLC) | Part 2D: BMS-986218 + Nivolumab Microsatellite Stable Colorectal Cancer (MSS CRC)
Number analyzed (Participants) | 2 | 4 | 5 | 3 | 4 | 1 | 2 | 4 | 0 | 2 | 1 | 1 | 0 | 2 | 3 | 5 | 1 | 0 | 10 | 8 | 6 | 7 | 10 | 10 | 11 | 9
hour | 233.28 (50.61) | 264.58 (16.51) | 274.01 (23.40) | 191.02 (19.95) | 175.33 (34.46) | 331.17 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 290.94 (6.57) | 234.91 (23.01) |  | 191.02 (4.42) | 200.61 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 211.88 (NA) — Insufficient number of participants to calculate geometric coefficient of variation |  | 213.34 (4.94) | 203.14 (2.92) | 205.63 (25.20) | 194.21 (NA) — Insufficient number of participants to calculate geometric coefficient of variation |  | 224.90 (33.11) | 271.49 (24.13) | 207.59 (16.53) | 233.09 (11.04) | 230.66 (32.95) | 235.80 (23.08) | 201.22 (41.29) | 198.93 (32.68)

21. Secondary Outcome: Time of Maximum Observed Concentration (Tmax) for BMS-986218
Description: Tmax is the time taken to reach the maximum observed serum concentration (Cmax) for BMS-986218.
Time Frame: On Cycle 1 Day 1, Cycle 1 Day 15, Cycle 3 Day 1, Cycle 3 Day 15 (Each Cycle is of 28 Days)
Population: All PK participants with available PK results at each time point
Measure: Median (Full Range); unit: hour
Arm/Group | Part 1A: BMS-986218 2 mg All Solid Tumors | Part 1A: BMS-986218 4 mg All Solid Tumors | Part 1A: BMS-986218 7 mg All Solid Tumors | Part 1A: BMS-986218 20 mg All Solid Tumors | Part 1A: BMS-986218 40 mg All Solid Tumors | Part 1A: BMS-986218 70 mg All Solid Tumors | Part 1A: BMS-986218 100 mg All Solid Tumors | Part 1A: BMS-986218 150 mg All Solid Tumors | Part 1A: BMS-986218 200 mg All Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors | Part 1A: BMS-986218 35 mg Select Solid Tumors | Part 1A: BMS-986218 50 mg Select Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors Pharmacodynamics Cohort | Part 1B: BMS-986218 7 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 20 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 40 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 70 mg + Nivolumab 480 mg Select Solid Tumors | Part 2A: Ipilimumab Cutaneous Melanoma | Part 2A: BMS-986218 7 mg Cutaneous Melanoma | Part 2A: BMS-986218 20 mg Cutaneous Melanoma | Part 2A: BMS-986218 70 mg Cutaneous Melanoma | Part 2B: BMS-986218 7 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 20 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 70 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2C: BMS-986218 + Nivolumab Non-Small Cell Lung Cancer (NSCLC) | Part 2D: BMS-986218 + Nivolumab Microsatellite Stable Colorectal Cancer (MSS CRC)
Number analyzed (Participants) | 4 | 9 | 12 | 15 | 12 | 14 | 7 | 11 | 5 | 14 | 6 | 4 | 1 | 5 | 17 | 18 | 7 | 0 | 15 | 17 | 17 | 20 | 20 | 20 | 27 | 41
hour
  Cycle 1 Day 1 | 2.04 [0.07 to 168.08] | 0.35 [0.13 to 4.13] | 0.48 [0.23 to 4.00] | 0.53 [0.47 to 24.58] | 0.52 [0.42 to 0.60] | 0.54 [0.47 to 24.00] | 0.70 [0.52 to 24.83] | 0.53 [0.47 to 25.08] | 0.60 [0.50 to 24.58] | 0.56 [0.50 to 21.87] | 11.51 [0.47 to 24.52] | 0.53 [0.50 to 0.58] | 20.93 [20.93 to 20.93] | 0.27 [0.12 to 24.23] | 0.52 [0.47 to 24.07] | 0.60 [0.47 to 166.17] | 0.62 [0.35 to 24.43] |  | 0.30 [0.23 to 24.35] | 0.58 [0.47 to 166.58] | 0.58 [0.47 to 24.25] | 0.27 [0.20 to 24.32] | 9.88 [0.42 to 162.42] | 0.53 [0.03 to 25.30] | 0.65 [0.50 to 22.50] | 0.92 [0.50 to 72.93]
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 15 |  |  |  |  |  |  |  |  |  | 0.52 [0.48 to 44.73] | 12.28 [0.50 to 25.72] | 12.15 [0.53 to 24.18] |  |  |  |  |  |  |  |  |  |  |  |  |  |
  Cycle 3 Day 1: number analyzed (Participants) | 2 | 4 | 6 | 4 | 4 | 2 | 3 | 4 | 0 | 3 | 2 | 2 | 1 | 2 | 4 | 7 | 1 | 0 | 13 | 12 | 8 | 11 | 12 | 10 | 11 | 9
  Cycle 3 Day 1 | 2.05 [0.10 to 4.00] | 2.08 [0.10 to 4.00] | 0.48 [0.25 to 4.33] | 12.24 [0.50 to 24.00] | 0.51 [0.42 to 0.53] | 0.68 [0.55 to 0.82] | 0.50 [0.50 to 0.70] | 0.53 [0.52 to 24.50] |  | 0.53 [0.47 to 0.53] | 12.41 [0.82 to 24.00] | 0.64 [0.53 to 0.75] | 0.52 [0.52 to 0.52] | 0.33 [0.25 to 0.40] | 21.06 [0.52 to 24.62] | 0.53 [0.47 to 21.82] | 0.75 [0.75 to 0.75] |  | 0.27 [0.20 to 24.00] | 0.53 [0.50 to 24.00] | 0.53 [0.47 to 167.92] | 0.28 [0.23 to 164.97] | 0.56 [0.47 to 24.60] | 0.52 [0.47 to 24.50] | 0.68 [0.00 to 24.00] | 0.75 [0.50 to 4.92]
  Cycle 3 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 3 Day 15 |  |  |  |  |  |  |  |  |  | 0.53 [0.53 to 0.53] | 12.26 [0.52 to 24.00] | 0.53 [0.53 to 0.53] | 0.53 [0.53 to 0.53] |  |  |  |  |  |  |  |  |  |  |  |  |

22. Secondary Outcome: Trough Observed Plasma Concentration (Ctrough) for BMS-986218
Description: Ctrough is the lowest observed serum concentration for BMS-986218.
Time Frame: At Cycle 1 Day 15, Cycle 2 Day 1, Cycle 2 Day 15, Cycle 3 Day 1, Cycle 3 Day 15, Cycle 4 Day 1, Cycle 5 Day 1, Cycle 7 Day 1, Cycle 9 Day 1, Cycle 13 Day 1, Cycle 17 Day 1, Cycle 21 Day 1 (Each Cycle is of 28 Days)
Population: All PK participants with available PK results at each time point
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Part 1A: BMS-986218 2 mg All Solid Tumors | Part 1A: BMS-986218 4 mg All Solid Tumors | Part 1A: BMS-986218 7 mg All Solid Tumors | Part 1A: BMS-986218 20 mg All Solid Tumors | Part 1A: BMS-986218 40 mg All Solid Tumors | Part 1A: BMS-986218 70 mg All Solid Tumors | Part 1A: BMS-986218 100 mg All Solid Tumors | Part 1A: BMS-986218 150 mg All Solid Tumors | Part 1A: BMS-986218 200 mg All Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors | Part 1A: BMS-986218 35 mg Select Solid Tumors | Part 1A: BMS-986218 50 mg Select Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors Pharmacodynamics Cohort | Part 1B: BMS-986218 7 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 20 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 40 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 70 mg + Nivolumab 480 mg Select Solid Tumors | Part 2A: Ipilimumab Cutaneous Melanoma | Part 2A: BMS-986218 7 mg Cutaneous Melanoma | Part 2A: BMS-986218 20 mg Cutaneous Melanoma | Part 2A: BMS-986218 70 mg Cutaneous Melanoma | Part 2B: BMS-986218 7 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 20 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 70 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2C: BMS-986218 + Nivolumab Non-Small Cell Lung Cancer (NSCLC) | Part 2D: BMS-986218 + Nivolumab Microsatellite Stable Colorectal Cancer (MSS CRC)
Number analyzed (Participants) | 3 | 6 | 9 | 7 | 8 | 5 | 3 | 4 | 3 | 10 | 4 | 4 | 1 | 5 | 11 | 9 | 5 | 0 | 14 | 13 | 13 | 17 | 16 | 15 | 21 | 24
ng/ml
  Cycle 1 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 15 |  |  |  |  |  |  |  |  |  | 751.99 (42.10) | 1501.35 (32.91) | 2793.34 (31.31) |  |  |  |  |  |  |  |  |  |  |  |  |  |
  Cycle 2 Day 1: number analyzed (Participants) | 3 | 6 | 9 | 7 | 8 | 5 | 3 | 4 | 3 | 9 | 3 | 4 | 0 | 5 | 11 | 9 | 5 | 0 | 14 | 13 | 13 | 17 | 16 | 15 | 21 | 24
  Cycle 2 Day 1 | 25.00 (0.00) | 55.05 (54.39) | 182.56 (59.17) | 341.81 (49.20) | 524.48 (65.16) | 1310.07 (42.38) | 1651.31 (39.58) | 2427.50 (68.46) | 2460.51 (38.43) | 1016.63 (57.51) | 1651.22 (51.66) | 3630.54 (21.56) |  | 99.96 (45.22) | 217.64 (62.28) | 466.94 (66.02) | 607.17 (75.73) |  | 129.05 (70.92) | 587.71 (143.00) | 1064.56 (48.39) | 141.23 (113.06) | 407.90 (62.10) | 1076.42 (60.99) | 423.18 (63.54) | 383.71 (71.78)
  Cycle 2 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 3 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 15 |  |  |  |  |  |  |  |  |  | 1063.74 (53.79) | 1547.03 (61.55) | 3029.39 (57.40) | 1450.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation |  |  |  |  |  |  |  |  |  |  |  |  |
  Cycle 3 Day 1: number analyzed (Participants) | 2 | 4 | 6 | 4 | 4 | 2 | 3 | 4 | 0 | 3 | 2 | 2 | 1 | 2 | 4 | 7 | 1 | 0 | 11 | 11 | 8 | 11 | 12 | 8 | 11 | 9
  Cycle 3 Day 1 | 41.86 (67.07) | 66.16 (45.96) | 297.97 (123.19) | 457.55 (55.91) | 229.14 (72.40) | 2337.71 (14.44) | 1260.06 (65.56) | 3163.13 (56.11) |  | 1174.88 (44.26) | 1266.41 (105.11) | 2637.27 (33.60) | 1860.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 59.16 (98.57) | 191.74 (68.64) | 356.38 (54.16) | 319.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation |  | 158.43 (77.94) | 459.88 (79.40) | 961.90 (41.84) | 224.06 (49.56) | 455.88 (69.43) | 1721.74 (44.78) | 532.21 (192.34) | 346.90 (55.72)
  Cycle 3 Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 3 Day 15 |  |  |  |  |  |  |  |  |  | 1273.50 (25.66) | 2723.07 (23.06) | 1930.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 1550.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation |  |  |  |  |  |  |  |  |  |  |  |  |
  Cycle 4 Day 1: number analyzed (Participants) | 1 | 3 | 4 | 1 | 2 | 1 | 1 | 2 | 0 | 1 | 2 | 0 | 0 | 2 | 4 | 5 | 1 | 0 | 8 | 6 | 3 | 6 | 6 | 8 | 7 | 6
  Cycle 4 Day 1 | 76.30 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 65.16 (60.55) | 239.17 (42.21) | 149.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 119.37 (129.54) | 2310.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 2650.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 5028.98 (43.48) |  | 1980.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 3212.85 (27.42) |  |  | 140.76 (67.67) | 159.03 (70.17) | 592.11 (63.58) | 339.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation |  | 190.56 (64.87) | 536.11 (51.32) | 850.80 (10.98) | 179.31 (37.25) | 579.85 (57.85) | 1473.97 (45.56) | 365.27 (102.58) | 734.46 (37.26)
  Cycle 5 Day 1: number analyzed (Participants) | 1 | 2 | 4 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 6 | 5 | 2 | 3 | 3 | 6 | 4 | 3
  Cycle 5 Day 1 | 57.70 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 76.43 (45.86) | 219.06 (30.71) | 155.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 243.09 (36.27) |  |  |  |  | 1890.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 3840.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation |  |  | 255.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 448.60 (8.97) | 1013.99 (84.49) |  |  | 209.59 (52.65) | 704.66 (24.65) | 1902.00 (31.19) | 108.85 (49.50) | 460.96 (112.61) | 1462.14 (44.11) | 318.78 (94.16) | 518.96 (71.39)
  Cycle 7 Day 1: number analyzed (Participants) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 7 Day 1 | 80.30 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 46.34 (77.66) |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |
  Cycle 9 Day 1: number analyzed (Participants) | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1
  Cycle 9 Day 1 |  | 85.46 (61.35) | 356.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation |  | 196.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation |  |  |  |  | 1710.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation |  |  |  | 232.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation |  |  |  |  | 570.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 770.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 932.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 123.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 2030.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 2110.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation |  | 646.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation
  Cycle 13 Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 1
  Cycle 13 Day 1 |  | 67.50 (NA) — Insufficient number of participants to calculate geometric coefficient of variation |  |  | 891.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation |  |  |  |  |  |  |  |  |  |  |  |  |  | 533.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 706.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 1020.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 203.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation |  | 1470.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation |  | 1820.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation
  Cycle 17 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1
  Cycle 17 Day 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 335.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation | 357.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation |  | 231.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation |  | 1150.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation |  | 1600.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation
  Cycle 21 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Cycle 21 Day 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 169.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation |  | 715.00 (NA) — Insufficient number of participants to calculate geometric coefficient of variation |  |

23. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA) to BMS-986218
Description: Baseline ADA Positive: Participant with baseline ADA-positive sample
  ADA Positive: Participant with at least one ADA-positive sample relative to baseline (ADA negative at baseline or ADA titer to be at least 4-fold or greater (>=) than baseline positive titer) at any time after initiation of treatment
  Persistent Positive (PP): ADA-positive sample at 2 or more consecutive timepoints, where the first and last ADA-positive samples are at least 16weeks apart
  Not PP-Last Sample Positive: Not persistent but with ADA-positive sample at the last sampling timepoint
  Other Positive: Not persistent but some ADA-positive samples with the last sample being negative
  ADA Negative: Participant with no ADA-positive sample after initiation of treatment
Time Frame: as for outcome 1
Population: All Treated Participants with BMS-986128 Who have Baseline and at Least One Post-baseline Pre-infusion ADA Assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: BMS-986218 2 mg All Solid Tumors | Part 1A: BMS-986218 4 mg All Solid Tumors | Part 1A: BMS-986218 7 mg All Solid Tumors | Part 1A: BMS-986218 20 mg All Solid Tumors | Part 1A: BMS-986218 40 mg All Solid Tumors | Part 1A: BMS-986218 70 mg All Solid Tumors | Part 1A: BMS-986218 100 mg All Solid Tumors | Part 1A: BMS-986218 150 mg All Solid Tumors | Part 1A: BMS-986218 200 mg All Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors | Part 1A: BMS-986218 35 mg Select Solid Tumors | Part 1A: BMS-986218 50 mg Select Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors Pharmacodynamics Cohort | Part 1B: BMS-986218 7 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 20 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 40 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 70 mg + Nivolumab 480 mg Select Solid Tumors | Part 2A: Ipilimumab Cutaneous Melanoma | Part 2A: BMS-986218 7 mg Cutaneous Melanoma | Part 2A: BMS-986218 20 mg Cutaneous Melanoma | Part 2A: BMS-986218 70 mg Cutaneous Melanoma | Part 2B: BMS-986218 7 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 20 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 70 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2C: BMS-986218 + Nivolumab Non-Small Cell Lung Cancer (NSCLC) | Part 2D: BMS-986218 + Nivolumab Microsatellite Stable Colorectal Cancer (MSS CRC)
Number analyzed (Participants) | 4 | 7 | 10 | 13 | 9 | 10 | 4 | 7 | 5 | 8 | 5 | 3 | 0 | 4 | 12 | 11 | 6 | 0 | 18 | 14 | 11 | 19 | 19 | 17 | 20 | 26
Participants
  Baseline ADA Positive | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 |  | 0 | 0 | 0 | 0 |  | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  ADA Positive | 0 | 1 | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 1 | 0 | 1 |  | 0 | 2 | 0 | 0 |  | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
  ADA Positive [Persistent Positive (PP)] | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ADA Positive [Not PP-Last Sample Positive] | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 |  | 0 | 2 | 0 | 0 |  | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  ADA Positive [Other Positive] | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 |  | 0 | 0 | 0 | 0 |  | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  ADA Negative | 4 | 6 | 10 | 12 | 9 | 7 | 3 | 7 | 5 | 7 | 5 | 2 |  | 4 | 10 | 11 | 6 |  | 18 | 13 | 10 | 19 | 18 | 17 | 20 | 26

ADVERSE EVENTS:
Time Frame: Participants were assessed for All-Cause Mortality from the date of their randomization (Part 2A and 2B) or first dose (Part 1, 2C and 2D) until study completion (assessed up to approximately 83 months). SAEs and Other AEs were assessed from first dose of study medication through 100 days following last dose of study treatment (assessed for an average of 8 months up to a max of approximately 28 months).
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants (Part 2A and 2B) or all participants that received at least 1 dose of study medication (Part 1, 2C and 2D).
  Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Arm/Group | Part 1A: BMS-986218 2 mg All Solid Tumors | Part 1A: BMS-986218 4 mg All Solid Tumors | Part 1A: BMS-986218 7 mg All Solid Tumors | Part 1A: BMS-986218 20 mg All Solid Tumors | Part 1A: BMS-986218 40 mg All Solid Tumors | Part 1A: BMS-986218 70 mg All Solid Tumors | Part 1A: BMS-986218 100 mg All Solid Tumors | Part 1A: BMS-986218 150 mg All Solid Tumors | Part 1A: BMS-986218 200 mg All Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors | Part 1A: BMS-986218 35 mg Select Solid Tumors | Part 1A: BMS-986218 50 mg Select Solid Tumors | Part 1A: BMS-986218 20 mg Select Solid Tumors Pharmacodynamics Cohort | Part 1B: BMS-986218 7 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 20 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 40 mg + Nivolumab 480 mg Select Solid Tumors | Part 1B: BMS-986218 70 mg + Nivolumab 480 mg Select Solid Tumors | Part 2A: Ipilimumab Cutaneous Melanoma | Part 2A: BMS-986218 7 mg Cutaneous Melanoma | Part 2A: BMS-986218 20 mg Cutaneous Melanoma | Part 2A: BMS-986218 70 mg Cutaneous Melanoma | Part 2B: BMS-986218 7 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 20 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2B: BMS-986218 70 mg Non-Small Cell Lung Cancer (NSCLC) | Part 2C: BMS-986218 + Nivolumab Non-Small Cell Lung Cancer (NSCLC) | Part 2D: BMS-986218 + Nivolumab Microsatellite Stable Colorectal Cancer (MSS CRC)
All-Cause Mortality (participants affected / at risk) | 2/4 | 7/9 | 6/12 | 10/15 | 8/12 | 7/14 | 6/7 | 10/11 | 1/5 | 9/14 | 6/6 | 3/4 | 1/1 | 4/5 | 15/17 | 14/19 | 5/7 | 13/20 | 16/19 | 16/18 | 18/18 | 19/22 | 20/22 | 16/22 | 28/29 | 37/44
Serious Adverse Events (participants affected / at risk) | 2/4 | 5/9 | 5/12 | 9/15 | 10/12 | 7/14 | 5/7 | 7/11 | 5/5 | 10/14 | 4/6 | 3/4 | 1/1 | 3/5 | 13/17 | 18/19 | 7/7 | 9/20 | 11/19 | 12/18 | 12/18 | 16/22 | 15/22 | 17/22 | 23/29 | 34/44
Other Adverse Events (participants affected / at risk) | 4/4 | 9/9 | 11/12 | 15/15 | 11/12 | 14/14 | 7/7 | 11/11 | 5/5 | 13/14 | 5/6 | 4/4 | 1/1 | 5/5 | 16/17 | 19/19 | 7/7 | 18/20 | 19/19 | 15/18 | 16/18 | 21/22 | 21/22 | 21/22 | 27/29 | 43/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A: BMS-986218 2 mg All Solid Tumors (N=4) | Part 1A: BMS-986218 4 mg All Solid Tumors (N=9) | Part 1A: BMS-986218 7 mg All Solid Tumors (N=12) | Part 1A: BMS-986218 20 mg All Solid Tumors (N=15) | Part 1A: BMS-986218 40 mg All Solid Tumors (N=12) | Part 1A: BMS-986218 70 mg All Solid Tumors (N=14) | Part 1A: BMS-986218 100 mg All Solid Tumors (N=7) | Part 1A: BMS-986218 150 mg All Solid Tumors (N=11) | Part 1A: BMS-986218 200 mg All Solid Tumors (N=5) | Part 1A: BMS-986218 20 mg Select Solid Tumors (N=14) | Part 1A: BMS-986218 35 mg Select Solid Tumors (N=6) | Part 1A: BMS-986218 50 mg Select Solid Tumors (N=4) | Part 1A: BMS-986218 20 mg Select Solid Tumors Pharmacodynamics Cohort (N=1) | Part 1B: BMS-986218 7 mg + Nivolumab 480 mg Select Solid Tumors (N=5) | Part 1B: BMS-986218 20 mg + Nivolumab 480 mg Select Solid Tumors (N=17) | Part 1B: BMS-986218 40 mg + Nivolumab 480 mg Select Solid Tumors (N=19) | Part 1B: BMS-986218 70 mg + Nivolumab 480 mg Select Solid Tumors (N=7) | Part 2A: Ipilimumab Cutaneous Melanoma (N=20) | Part 2A: BMS-986218 7 mg Cutaneous Melanoma (N=19) | Part 2A: BMS-986218 20 mg Cutaneous Melanoma (N=18) | Part 2A: BMS-986218 70 mg Cutaneous Melanoma (N=18) | Part 2B: BMS-986218 7 mg Non-Small Cell Lung Cancer (NSCLC) (N=22) | Part 2B: BMS-986218 20 mg Non-Small Cell Lung Cancer (NSCLC) (N=22) | Part 2B: BMS-986218 70 mg Non-Small Cell Lung Cancer (NSCLC) (N=22) | Part 2C: BMS-986218 + Nivolumab Non-Small Cell Lung Cancer (NSCLC) (N=29) | Part 2D: BMS-986218 + Nivolumab Microsatellite Stable Colorectal Cancer (MSS CRC) (N=44)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immune-mediated myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 5 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 3 | 0 | 1
Duodenal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 5 | 1 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Malignant ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pancreatic mass (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 5
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Immune-mediated cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sarcoidosis (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess soft tissue (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Biliary sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Biliary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis intestinal perforated (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis yersinia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematological infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Norovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 1 | 1
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stoma prolapse (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin T increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1 | 2 | 3 | 2 | 2 | 4 | 1 | 6 | 3 | 1 | 0 | 2 | 8 | 8 | 2 | 1 | 3 | 6 | 6 | 8 | 9 | 3 | 10 | 13
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour fistulisation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immune-mediated encephalitis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intracranial tumour haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device dislocation (Product Issues) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 3 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A: BMS-986218 2 mg All Solid Tumors (N=4) | Part 1A: BMS-986218 4 mg All Solid Tumors (N=9) | Part 1A: BMS-986218 7 mg All Solid Tumors (N=12) | Part 1A: BMS-986218 20 mg All Solid Tumors (N=15) | Part 1A: BMS-986218 40 mg All Solid Tumors (N=12) | Part 1A: BMS-986218 70 mg All Solid Tumors (N=14) | Part 1A: BMS-986218 100 mg All Solid Tumors (N=7) | Part 1A: BMS-986218 150 mg All Solid Tumors (N=11) | Part 1A: BMS-986218 200 mg All Solid Tumors (N=5) | Part 1A: BMS-986218 20 mg Select Solid Tumors (N=14) | Part 1A: BMS-986218 35 mg Select Solid Tumors (N=6) | Part 1A: BMS-986218 50 mg Select Solid Tumors (N=4) | Part 1A: BMS-986218 20 mg Select Solid Tumors Pharmacodynamics Cohort (N=1) | Part 1B: BMS-986218 7 mg + Nivolumab 480 mg Select Solid Tumors (N=5) | Part 1B: BMS-986218 20 mg + Nivolumab 480 mg Select Solid Tumors (N=17) | Part 1B: BMS-986218 40 mg + Nivolumab 480 mg Select Solid Tumors (N=19) | Part 1B: BMS-986218 70 mg + Nivolumab 480 mg Select Solid Tumors (N=7) | Part 2A: Ipilimumab Cutaneous Melanoma (N=20) | Part 2A: BMS-986218 7 mg Cutaneous Melanoma (N=19) | Part 2A: BMS-986218 20 mg Cutaneous Melanoma (N=18) | Part 2A: BMS-986218 70 mg Cutaneous Melanoma (N=18) | Part 2B: BMS-986218 7 mg Non-Small Cell Lung Cancer (NSCLC) (N=22) | Part 2B: BMS-986218 20 mg Non-Small Cell Lung Cancer (NSCLC) (N=22) | Part 2B: BMS-986218 70 mg Non-Small Cell Lung Cancer (NSCLC) (N=22) | Part 2C: BMS-986218 + Nivolumab Non-Small Cell Lung Cancer (NSCLC) (N=29) | Part 2D: BMS-986218 + Nivolumab Microsatellite Stable Colorectal Cancer (MSS CRC) (N=44)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 3 | 4 | 4 | 2 | 3 | 2 | 4 | 7 | 1 | 0 | 0 | 3 | 4 | 3 | 6 | 6 | 8 | 8 | 3 | 4 | 4 | 12 | 9 | 20
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 2 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Glucocorticoid deficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 3 | 4
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 5
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Exophthalmos (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye inflammation (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital swelling (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 2 | 2 | 1 | 2 | 0 | 3 | 1 | 5 | 1 | 1 | 0 | 0 | 4 | 4 | 0 | 2 | 2 | 2 | 2 | 1 | 3 | 5 | 5 | 11
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 4 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 7 | 4 | 3 | 2 | 1 | 2 | 1 | 7 | 0 | 0 | 0 | 2 | 3 | 3 | 0 | 1 | 5 | 4 | 4 | 1 | 4 | 2 | 5 | 9
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 5 | 4 | 3 | 3 | 3 | 3 | 4 | 1 | 3 | 0 | 0 | 3 | 5 | 5 | 7 | 8 | 4 | 7 | 3 | 5 | 9 | 9 | 16
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 3
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gingival swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 3 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 0 | 4 | 0 | 3 | 2 | 3 | 3 | 5 | 0 | 0 | 0 | 1 | 6 | 5 | 2 | 5 | 5 | 4 | 2 | 2 | 4 | 5 | 10 | 17
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Rectal discharge (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4
Tongue oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 4 | 1 | 3 | 1 | 2 | 2 | 0 | 2 | 4 | 0 | 0 | 0 | 2 | 4 | 4 | 0 | 3 | 1 | 3 | 1 | 2 | 2 | 4 | 6 | 10
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 6 | 0 | 5 | 3 | 2 | 2 | 2 | 1 | 4 | 3 | 8
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 3 | 2 | 6 | 3 | 7 | 3 | 7 | 1 | 5 | 3 | 0 | 0 | 1 | 9 | 9 | 5 | 3 | 6 | 7 | 4 | 5 | 11 | 10 | 12 | 19
Gait disturbance (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 2 | 1 | 1 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1 | 3 | 3 | 1 | 1 | 4 | 2 | 4 | 1 | 0 | 0 | 1 | 2 | 2 | 3 | 2 | 1 | 0 | 1 | 4 | 0 | 1 | 4 | 5
Pain (General disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 4 | 3 | 2 | 1 | 4 | 3 | 0 | 2 | 2 | 0 | 0 | 2 | 9 | 4 | 2 | 2 | 1 | 3 | 0 | 2 | 6 | 4 | 19
Xerosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Biliary dilatation (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rubber sensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sarcoidosis (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Biliary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 5
Candida infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 1
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea cruris (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 2 | 1 | 2 | 1 | 2 | 1 | 2 | 0 | 4
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 6
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Vascular access site erythema (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular access site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 2 | 1 | 2 | 1 | 2 | 0 | 3 | 1 | 0 | 0 | 0 | 1 | 5 | 3 | 4 | 2 | 3 | 3 | 1 | 5 | 3 | 4 | 14
Amylase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 4 | 1 | 3 | 1 | 2 | 2 | 1 | 6
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 2 | 2 | 2 | 1 | 1 | 1 | 3 | 1 | 0 | 0 | 2 | 2 | 7 | 4 | 3 | 4 | 3 | 2 | 1 | 4 | 3 | 5 | 12
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 1 | 1 | 2 | 4
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 0 | 2 | 0 | 3 | 0 | 2 | 2 | 2 | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 6
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 1 | 1 | 3 | 0 | 1 | 1 | 2 | 2 | 0 | 0 | 1 | 1 | 3 | 2 | 1 | 2 | 1 | 2 | 0 | 1 | 1 | 1 | 12
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 1
Blood calcium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 0 | 0 | 1 | 0 | 2 | 1
Blood creatinine increased (Investigations) | 1 | 3 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 3 | 0 | 4 | 0 | 2 | 1 | 1 | 5 | 6
Blood fibrinogen decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 2 | 2 | 0 | 0 | 3
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 0 | 0 | 2 | 2 | 3 | 6
Blood magnesium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 4 | 0 | 2 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0
Eosinophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fibrin D dimer increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 4
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lipase increased (Investigations) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 4 | 1 | 3 | 2 | 1 | 3 | 5 | 9
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 2
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Platelet count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 2
Troponin T increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Viral test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 1 | 1 | 1 | 2 | 0 | 0 | 1 | 7 | 4 | 2 | 0 | 1 | 1 | 2 | 1 | 1 | 5 | 2 | 5
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 0 | 4 | 2 | 1 | 1 | 7 | 2 | 2 | 1 | 0 | 0 | 0 | 6 | 11 | 2 | 3 | 4 | 3 | 2 | 5 | 10 | 8 | 8 | 16
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 3 | 2
Folate deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 2 | 4 | 3 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 3 | 3 | 2 | 0 | 0 | 0 | 1 | 1 | 2 | 3 | 1 | 3 | 0 | 1 | 1 | 0 | 2 | 1 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 3 | 4 | 3 | 1 | 0 | 0 | 0 | 2 | 4 | 1 | 1 | 4 | 2 | 3 | 2 | 0 | 2 | 4 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 2 | 1 | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 3 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 1 | 4 | 3 | 1 | 4 | 4 | 4 | 0 | 0 | 0 | 1 | 4 | 3 | 3 | 3 | 3 | 2 | 1 | 1 | 0 | 4 | 4 | 7
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 2 | 1 | 2 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 2
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Steroid diabetes (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 4 | 1 | 2 | 1 | 1 | 4 | 1 | 0 | 0 | 1 | 0 | 4 | 2 | 0 | 0 | 2 | 2 | 3 | 0 | 2 | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3 | 2 | 2 | 4 | 2 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 3 | 0 | 1 | 0 | 1 | 2 | 2 | 4 | 1 | 1 | 1 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mandibular mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1 | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 3 | 1 | 0 | 2 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cauda equina syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 2
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 2
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 3 | 2 | 2 | 0 | 2 | 4 | 3 | 3 | 1 | 4 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intracranial tumour haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 3 | 1 | 0 | 1 | 1 | 4 | 2 | 3 | 4
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Persistent depressive disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pelvic haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Testicular disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Testicular oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 3 | 2 | 2 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 3 | 1 | 1 | 3 | 5 | 6 | 6 | 11
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 1 | 1 | 0 | 3 | 4 | 1 | 3 | 0 | 0 | 0 | 2 | 2 | 4 | 0 | 1 | 2 | 0 | 3 | 7 | 7 | 6 | 6 | 8
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Malignant pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 4 | 1 | 2 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 4 | 2 | 5 | 8 | 3 | 6 | 1 | 4 | 4 | 5 | 6
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 1 | 2 | 3 | 3 | 2 | 6
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 2 | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 2 | 0 | 1 | 2 | 2 | 3 | 0 | 6 | 4
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sensitive skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 5 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 3
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Superficial vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/07/NCT03110107/Prot_SAP_000.pdf